# Statistical Analysis Plan Part A and B

SAFETY AND IMMUNOGENICITY STUDY OF VLA15, A MULTIVALENT RECOMBINANT OSPA BASED VACCINE CANDIDATE AGAINST LYME BORRELIOSIS: A RANDOMIZED, CONTROLLED, OBSERVER-BLIND PHASE 2 STUDY IN A HEALTHY PEDIATRIC AND ADULT STUDY POPULATION

Protocol: VLA15-221

Confidential

Study Sponsor: Pfizer

Study Conducted By: Valneva Austria GmbH

# **Table of Contents**

| 1. | OVER | VIEW | 9 |
|---|---|---|---|
| | 1.1<br>1.1.1<br>1.1.2 | Study Objectives Primary Objective Secondary Objectives | 9<br>9<br>9 |
| | 1.2 | Study Design | 9 |
| | 1.3<br>1.3.1<br>1.3.2<br>1.3.3 | Endpoints Primary Endpoint Secondary Endpoints Exploratory endpoints | 12<br>12<br>12<br>13 |
| | 1.4 | Sample Size Calculation | 13 |
| | 1.5<br>1.5.1<br>1.5.2 | Flowchart Study Design Study Schedule | 14<br>14<br>15 |
| 2. | GENE | RAL CONSIDERATIONS | 19 |
| | 2.1 | Conduct of Analysis | 19 |
| | 2.2 | Statistical Software and Quality Control | 19 |
| | 2.3 | Applicable Standard Operating Procedures | 20 |
| | 2.4 | Randomization and Blinding | 20 |
| | 2.5 | Descriptive Analyses | 21 |
| | 2.6 | Center and Country Effect and Stratification | 21 |
| | 2.7 | Handling Missing Data | 21 |
| | 2.8<br>2.8.1<br>2.8.2 | Protocol Deviations Part A: Main Study Phase Part B: Booster Phase | 22<br>22<br>22 |
| | 2.9 | Exclusion of Time Points in the Per-Protocol Analysis | 22 |
| | 2.10<br>2.10.1<br>2.10.2<br>2.10.3<br>2.10.4<br>2.10.5<br>2.10.6 | Full Analysis Set (FAS) Per-Protocol Analysis Set (PPAS) Booster Safety Analysis Set (BSAS) Booster Full Analysis Set (BFAS) | 23<br>23<br>24<br>24<br>24<br>24 |
| | 2.11 | Subject Data Listings | 24 |
| | 2.12 | Columns in Tables and Derivation of Actual Treatment | 24 |
| | 2.13 | Medical Coding | 26 |
| | 2.14 | Labelling of Visits | 26 |
| | 2.15 | Changes in the Conduct of the Study or Planned Analysis | 26 |
| | 2.16 | Effect of COVID-19 | 26 |
| 3. | OVER | ALL STUDY INFORMATION | 27 |

| | 3.1 | Data Points | 27 |
|---|---|---|---|
| | 3.2 | Definitions | 27 |
| 4. | BASE | LINE EVALUATION | 28 |
| | 4.1 | Data Points | 28 |
| | 4.2 | Definitions | 28 |
| 5. | IMMU | JNOGENICITY ANALYSIS | 29 |
| | 5.1<br>5.1.1<br>5.1.2 | Data Points Tables and Listings Figures for ELISA COLUMN | 30<br>30<br>31 |
| | 5.2<br>5.2.1 | Derivations and Definitions ELISA | 33<br>33<br>33 |
| | 5.3 | Statistical Tests | 34 |
| 6. | SAFE | TY ANALYSIS | 36 |
| | 6.1 | Adverse Events Documentation of Adverse Events Data Points Derivations and Definitions 3.1 General Principles for Analysis of Adverse Event 3.2 Principles for Solicited Adverse Events 3.3 Principles for Unsolicited Adverse Events Confidence Intervals and Statistical Tests | 36<br>36<br>38<br>38<br>39<br>41<br>42 |
| | 6.2<br>6.2.1<br>6.2.2 | Lyme Borreliosis Screening Data Points Derivations and Definitions | 42<br>42<br>42 |
| | 6.3 | Other Safety Parameters | 43 |
| 7. | LIST ( | DF TABLES, DATA LISTINGS AND FIGURES | 44 |
| | 7.1.1<br>7.1.2<br>7.1.3<br>7.1.4<br>7.1.5 | List of Tables Overall Study Information Baseline Evaluation Immunogenicity Analysis Adverse Events Other Safety Analysis and B.b. s.l. Serostatus | 46<br>46<br>48<br>49<br>66<br>80 |
| | 7.2<br>7.2.1<br>7.2.2<br>7.2.3<br>7.2.4<br>7.2.5 | List of Data Listings Overall Study Information Baseline Evaluation Immunogenicity Analysis Adverse Events Other Safety Analysis and B.b. s.l. Serostatus | 81<br>81<br>84<br>86<br>87<br>93 |
| | 7.3<br>7.3.1<br>7.3.2 | List of Figures<br>Immunogenicity Analysis<br>Adverse Events | 94<br>94<br>109 |
| 8. | SHEL | LS OF TABLES, DATA LISTINGS AND FIGURES | 110 |

| | Do | ocument | |
|---|---|---|---|
| Study | VLA15-221 | | |
| Document | Statistical Analysis Plan (S | SAP) | |
| Version | FINAL 2.0 | | |
| Date | 03-Mar-2022 | | |
| | Revis | sion History | |
| Version | Date | | n for Revision |
| FINAL 1.0 | 03-Jan-2022 | First version; | |
| FINAL 2.0 | 03-Mar-2022 | handling of vaccinations (concomitant medications definitions enhanced to a (programming of data cut programming for immuno missing assessments for assignment rules for AE); programming added, as s Meeting Report; tables fo 12 added; specific figures changes/corrections in la | void any possibility of ambiguity -off, time window violation genicity samples, handling of AE, vaccination period rule for actual treatment group pecified in Blind Data Review r GMFRs as compared to Month s by age cohort added; Minor yout, spelling, headers, and onfidence intervals for GMTs in |
| | A | pproval | |
| Name | Role | Date | Signature |
| | | Author | |
| PPD | Senior Biostatistician | | |
| PPD | Lead Biostatistician | | |





| Pfizer Inc. | |
|-------------|------------------------------------------|
| PPD | Program Statistician for<br>Lyme Vaccine |

Any photocopies taken of this document are not authorized or version controlled.

# **List of Abbreviations**

| AE | Adverse Event |
|---------|-----------------------------------|
| AESI | Adverse Event of Special Interest |
| ANOVA | Analysis of Variance |
| approx. | Approximately |
| BDRM | Blinded Data Review Meeting |
| CRA | Clinical Research Associates |
| CRO | Clinical Research Organization |
| DRM | Data Review Meeting |
| DSMB | Data Safety Monitoring Board |
| e.g. | exempli gratia |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| ELISA | Enzyme-Linked Immunosorbent Assay |
| EP | Endpoint |
| ET | Early Termination |
| FAS | Full Analysis Set |
| GMT | Geometric Mean Titer |
| GMFR | Geometric Mean Fold Rise |
| HIV | Human Immunodeficiency Virus |
| i.e. | id est |
| IgG | Immunoglobulin G |
| IMP | Investigational Medicinal Product |
| IRC | Internal Review Committee |
| mL | Milliliter(s) |
| OspA | Outer surface protein A |
| PBS | Polymerase Chain Reaction |
| PCR | Phosphate Buffered Saline |
| PP | Per-Protocol |
| PPAS | Per-Protocol Analysis Set |
| SAS | Statistical Analysis Set |
| SAE | Serious Adverse Event |
| CCI | |
| SCR | Seroconversion Rate |
| SD | Standard Deviation |



| SOP | Standard Operating Procedure |
|-----|------------------------------|
| ST | Serotype |
| TLF | Table, Listing and Figure |
| Yrs | Years |

Adapted from:
STAT03\_A Statistical Analysis Plan
Version 6.0, Effective Date 16-Feb-2018

#### OVERVIEW

#### 1.1 Study Objectives

#### 1.1.1 Primary Objective

#### Safety:

• To assess the safety and tolerability profile of VLA15, applied in a three- or two dose primary immunization schedule (Month 0-2-6 or Month 0-6), in a healthy study population aged 5 to 65 years up to Day 208 (Month 7).

#### Immunogenicity:

• To assess the immune response to VLA15, applied in a three- or two dose primary immunization schedule (Month 0-2-6 or Month 0-6), in a healthy study population aged 5 to 65 years at Day 208 (Month 7).

#### 1.1.2 Secondary Objectives

#### Safety:

- To assess the safety and tolerability profile of VLA15, applied in a three- or two dose primary immunization schedule (Month 0-2-6 or Month 0-6), in a healthy study population aged 5 to 65 years, up to one year after the last primary vaccination (Month 18);
- To assess the safety and tolerability profile of a booster dose of VLA15, applied one year after completion of the primary immunization schedule (i.e. Month 18), up to three years after the booster (i.e. Month 54).

#### Immunogenicity:

- To assess the immune response to VLA15, applied in a three- or two dose primary immunization schedule (Month 0-2-6 or Month 0-6), in a healthy study population aged 5 to 65 years, up to one year after the last primary vaccination (Month 18);
- To assess the immune response to a booster dose of VLA15, applied one year after completion of the primary immunization schedule (i.e. Month 18), up to three years after the booster (Month 54).

#### Exploratory objective:

#### 1.2 Study Design

VLA15-221 is a randomized, observer-blind (subject, sponsor and investigator/ site staff involved in clinical evaluation of subjects are blinded), placebo controlled, multicenter Phase 2 study in healthy subjects aged 5 to 65 years. The study is conducted in two study parts (Part A: Main Study Phase, Part B: Booster Phase, see Figure 1). VLA15-221 is initiated with an age de-escalation of sentinel cohorts. Subject enrollment into Part A starts with the adult cohort that allows the generation and review of appropriate safety data before pediatric cohorts are initiated. In Part A (Main Study Phase) a total of approximately 600 subjects aged 5 to 65 years is randomized 1:1:1 into three study groups: Group 1 (approximately 200 subjects) receives three vaccinations of VLA15 at Month 0-2-6. Group 2 (approximately 200 subjects) receives two VLA15 vaccinations at Month 0-6 and a placebo injection at

Adapted from: STATO3\_A Statistical Analysis Plan Version 6.0, Effective Date 16-Feb-2018 

Month 2 in order to keep the blind. Group 3 (approximately 200 subjects) receives three placebo injections at Month 0-2-6. Randomization is stratified by three age cohorts (18-65 years [n=300], 12-17 years [n=150] and 5-11 years [n=150]).

In Part A, all subjects receive three intramuscularly vaccinations at Month 0-2-6 (i.e. Day 1-57-180). On Day 8/Visit 1A (i.e. 7 days after the first vaccination) a safety visit is performed (phone call for subjects aged 18-65, in-person visit for subjects aged 5-17 years). In-person visits are scheduled for all age cohorts one month after each vaccination. Blood samples for immunogenicity assessments are collected at the screening visit, Day 85, Day 180, Day 194 (in a subset of adult subjects), Day 208, Day 365/Month 12 and at Month 18.

Based on safety and immunogenicity data from Day 208/Visit 6 of Part A (i.e. 1 month after the third immunization), data are used to guide the decision for Part B booster.

In **Part B (Booster Phase)** all eligible subjects from the Group that received selected primary schedule in Part A (either Group 1 or 2) receive a booster dose of VLA15 at Month 18.

For safety comparison, placebo injections are administered to approximately 100 subjects, who were vaccinated in Part A according to the alternative vaccination schedule, (i.e. either Group 1 or 2 which received vaccinations according to the primary immunization schedule that is not selected for further vaccine development), and to approximately 100 subjects of Group 3. It is targeted to maintain the 2:1:1 age stratification (18-65 years, 12-17 years and 5-11 years) in all study groups. All subjects involved in Part B are followed-up for further 3 years (i.e. up to Month 54) with study visits at Months 19, 23, 26, 30, 36, 42, 48 and 54.

Table 1: Study Groups and Vaccinations

| | Study Group | Subjects | Age in years | Treatment | Vaccination<br>Schedule |
|---|---|---|---|---|---|
| ase | Group 1 | Total: 200<br>100<br>50<br>50 | 18-65<br>12-17<br>5-11 | VLA15 180 µg | Month 0-2-6 |
| Part A: Main Study Phase | Group 2 | Total: 200<br>100<br>50<br>50 | 18-65<br>12-17<br>5-11 | VLA15 180 μg<br>Placebo | Month 0-6<br>Month 2* |
| Part | Group 3 | Total: 200<br>100<br>50<br>50 | 18-65<br>12-17<br>5-11 | Placebo | Month 0-2-6 |
| ISe | Group 1 or 2:<br>Selected<br>Schedule | Total: 200<br>100<br>50<br>50 | 18-65<br>12-17<br>5-11 | VLA15 180 μg | Month 18 |
| Part B: Booster Phase | Group 1 or 2:<br>Alternative<br>Schedule | Total: 100<br>50<br>25<br>25 | 18-65<br>12-17<br>5-11 | Placebo | Month 18 |
| <u>o</u> | Group 3 | Total: 100<br>50<br>25<br>25 | 18-65<br>12-17<br>5-11 | Placebo | Month 18 |

<sup>\*</sup>In order to keep the blind, subjects assigned to Group 2 will receive a sham injection of placebo at Month 2.

#### 1.3 Endpoints

#### 1.3.1 Primary Endpoint

#### Safety:

• Frequency of solicited local and solicited systemic Adverse Events (AEs) within 7 days after each and any vaccination of the primary vaccination series (Part A).

#### Immunogenicity:

 Geometric Mean Titers (GMTs) for Immunoglobulin G (IgG) against each OspA serotype ST1 to ST6, determined by an IgG binding assay, at Day 208/Month 7 (Part A).

#### 1.3.2 Secondary Endpoints

#### Safety:

- Frequency of solicited local and solicited systemic AEs within 7 days after booster dose administration (Part B);
- Frequency of Serious Adverse Events (SAEs) during the entire study;
- Frequency of Adverse Events of Special Interest (AESIs) during the entire study;
- Frequency of unsolicited AEs within 28 days after each vaccination;
- Frequency of SAEs, AESIs, unsolicited and solicited AEs stratified by age cohort.

#### Immunogenicity:

- Part A Main Study Phase:
  - o GMTs for IgG against each OspA serotype (ST1 to ST6), determined by an IgG binding assay, at baseline (screening visit) and at Day 85, 180, 194<sup>1</sup>, 365 and Month 18;
  - Seroconversion Rate SCRs, definition see Section 5.2.1) for each OspA serotype specific IgG (ST1 to ST6), determined by an IgG binding assay, at Day 85, 180, 194<sup>1</sup>, 208, 365 and Month 18;
  - Geometric Mean of the fold rise (GMFRs as compared to baseline) for IgG against each OspA serotype (ST1 to ST6), determined by an IgG binding assay, at Day 85 and 208;
  - GMTs, SCRs and GMFRs for IgG against each OspA serotype (ST1 to ST6), determined by an IgG binding assay, at specified time-points, stratified by age cohort.
- Part B Booster Phase:
  - GMTs for IgG against each OspA serotype (ST1 to ST6), determined by an IgG binding assay, at Month 18, 19, 23, 26, 30, 36, 42, 48 and 54;
  - SCRs for each OspA serotype specific IgG (ST1 to ST6), determined by an IgG binding assay, at Month 18, 19, 23, 26, 30, 36, 42, 48 and 54;
  - GMFRs for IgG against each OspA serotype (ST1 to ST6), determined by an IgG binding assay, at Month 19;

<sup>&</sup>lt;sup>1</sup> Visit 5A/Day194 data will be available for a subset of approximately 150 adult subjects.



 GMTs, SCRs and GMFRs for IgG against each OspA serotype (ST1 to ST6), determined by an IgG binding assay, at specified time points, stratified by age cohort.

## 1.3.3 Exploratory endpoints



#### 1.4 Sample Size Calculation

The sample size has been chosen to allow detection of common AEs. A total of 400 subjects in the VLA15 groups (Group 1 and Group 2) will provide 95% confidence that an AE not seen in the study would have a true incidence of not more than 0.75% across all age cohorts. In addition, the overall group size for the two VLA15 study groups has been selected to provide a sufficient safety database and for determining the optimal vaccination schedule before advancing the vaccine candidate into Phase 3. Upon completion of the study, the total number of subjects exposed to the final dose as used for upcoming Phase 3 studies would be a minimum of approximately N=710. The database would, thus, allow 95% confidence that a given reaction would not be observed at a higher rate than 1:(710/3) rate, i.e. 0.4%, if it is not observed in the studies preceding Phase 3.

With respect to the primary endpoint, GMTs for ST1-6 specific IgGs on Day 208: In the absence of an established protective titer, sample size calculation is based on somewhat arbitrary differences in GMTs between VLA15 study groups to demonstrate which titer levels could be distinguished with the proposed sample size.

Titers observed in the primary endpoint immunogenicity analysis (i.e. Day 208; one month after third vaccination) of 86 subjects receiving 180  $\mu$ g of VLA15 in ongoing Phase 2 study VLA15-202 were used as basis: In the 180  $\mu$ g group (i.e. the dose chosen for further development of VLA15), an Enzyme-Linked Immunosorbent Assay (ELISA) GMT of 274.7 was observed for ST1 (i.e. the serotype with lowest titers) with a Standard Deviation (LOG10) of 0.53. A total of 180 subjects per group (assuming 10% of the 200 subjects per study group are excluded from the primary Per-Protocol (PP) analysis) will provide 80% power at a two-sided alpha level of 5% to distinguish a GMT of 274.7 in one study group from a putative higher GMT of 394.3 in the other study group.

The overall sample size of 200 subjects in the placebo group has been selected to allow for the internal validation of both safety and immunogenicity results.

For the Booster Phase (Part B) no formal sample size calculation has been performed. All subjects that were randomized into the study group that received vaccinations according to the selected immunization schedule (Group 1 or Group 2) and are eligible, are foreseen to participate in Part B, while a total of approximately 100 subjects from the VLA15 group that received vaccinations according to the alternative primary schedule (Group 1 or 2) and approximately 100 subjects from Group 3 will be included in Part B.

#### 1.5 Flowchart

#### 1.5.1 Study Design

Figure 1: Study Design



- \* For subjects enrolled in Part B only
- + Visit 5A to be performed in a subset of approx. 150 adult (18-65 years) subjects only

#### 1.5.2 Study Schedule

Table 2: Table of Events - Part A: Main Study Phase

| Visit | V0 (1) | V1 (2) | V1A (3) | V2 (4) | V3 (2) | V4 (4) | V5 (2) | V5A (5) | V6 (4) | V7 (4) | V8 (4) | Early<br>Termination<br>(4) (6) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Timing Day (D)<br>Month (M) | D-10 | D1 | D8 | D29<br>M1 | D57<br>M2 | D85<br>M3<br>V3 + 28d | D180<br>M6 | D194<br>M6.5<br>V5 + 14d | D208<br>M7<br>V5 + 28d | D365<br>M12 | D545<br>M18 | < V8 |
| Time windows (D) | -10 to 0 | 0 | +2 | +2/- 4 | +/- 4 | +/- 4 | +4/-28 | +/-2 | +2/- 4 | +/- 14 | +/- 14 | n/a |
| Visit type | In-person | In-person | In-person<br>or remotely | In-person<br>or remotely | In-person | In-person<br>or remotely | In-person | In-person<br>or remotely | In-person<br>or remotely | In-person<br>or remotely | In-person<br>or remotely | In-person<br>or remotely |
| Informed consent/assent (7) | X | | | | | | | | | | | |
| Inclusion/exclusion criteria | X | X<br>(Review) | | | | | | | | | | |
| Vaccination delay criteria | | X | | | X | | X | | | | | |
| Demographic data | X | | | | | | | | | | | |
| Medical history incl. vaccinations | X | X (8) | | | | | | | | | | |
| Concomitant medications/<br>treatments incl. vaccinations | X | X | X | X | X | x | Х | X | X | x | X | x |
| Physical examination, ECG (9) | X | | | | | | | | | | | |
| Vital signs (10) | X | X | | | X | | X | | | | | |
| Evaluation of oral body temperature | X | X (11) | | | X (11) | | X (11) | | | | | |
| HIV test [3.0 mL] (12) | X | | | | | | | | | | | |
| B.b. s.l. screening test [5.0 mL] (13) | X | | | | | | | | | | X | X (14) |
| Serum Pregnancy test [2.0 mL] (15) | X | | | | | | | | | | | |
| Urine Pregnancy test (15) | | X (16) | | X | X (16) | X | X (16) | | X | X | X | X |
| Immunogenicity blood sample<br>[12.0 mL] (17) | X | | | | | X | X | Х | X | X | Х | |
| Assay development sample<br>[75.0 mL] (18) | | X | | | | x | | | X | | | |
| Randomization (19) | | X | | | | | | | | | | |
| VACCINATION (20) | | X | | | X | | X | | | | | |
| Check for AEs following vaccination | | X (21) | | | X (21) | | X (21) | | | | | |
| Symptom-driven physical exam (22) | | X | X (23) | X | X | X | X | X | X | X | X | X |
| Inspection of injection site of previous vaccinations | | | X (23) | X | | X | | Х | Х | | | X (25) |
| Explain eDiary (24) | | X | | | | | | | | | | |
| Review eDiary | | | X | X | | X | | X | X | | | X (26) |
| Check eDiary for SAEs/ AESIs | | | X | X | X | X | X | X | X | X | X | X |
| Scripted Safety Assessment | | | X | X | X | X | X | X | X | X | X | X |
| AE/ SAE/ AESI Assessment (27) | | | X | X | X | X | X | X | X | X | X | X |
| Blood Volume [mL] | 17.0 (28);<br>19.0 (29);<br>20.0 (30);<br>22.0 (31) | 75.0 (32) | 0.0 | 0.0 | 0.0 | 12.0 (33);<br>87.0 (34) | 12.0 | 12.0 | 12.0 (33);<br>87.0 (34) | 12.0 | 17.0 | 5.0 (14) |

Adapted from: STAT03\_A Statistical Analysis Plan Version 6.0, Effective Date 16-Feb-2018

without prior written consent of


Table 3: Table of Events - Part B. Booster Phase

| Visit | V8B (35) | V9 | V10 | V11 | V12 | V13 | V14 | V15 | V16 | Early<br>Termination (36) |
|---|---|---|---|---|---|---|---|---|---|---|
| Month (M) | M18 | M19<br>V8B + 28d | M23 | M26 | M30 | M36 | M42 | M48 | M54 | <v16< th=""></v16<> |
| Time windows (D) | V8 +14 | +/- 4 | +/- 14 | +/- 14 | +/-28 | +/-28 | +/-28 | +/-28 | +/-28 | n/a |
| Visit type | In-person | In-person | In-person | In-person | In-person | In-person | In-person | In-person | In-person | In-person |
| Inclusion/Exclusion criteria (Booster Phase) | X | | | | | | | | | |
| Vaccination delay criteria | X | | | | | | | | | |
| Concomitant medications/<br>treatments incl. vaccinations | X (37) | X | X | Х | Х | X | X | X | Х | х |
| Physical examination (9) | X | | | | | | | | | |
| Vital signs (10) | X | | | | | | | | | |
| Evaluation of oral body temperature | X (11) | | | | | | | | | |
| B.b. s.l. screening test [5.0 mL] (13) (38) | | | | | X | | X | | Х | Х |
| Urine Pregnancy test (15) | X (16) | X | X | | | | | | | X |
| Immunogenicity blood sample<br>[12.0 mL] (17) | | X | X | X | Х | X | X | X | X | |
| Assay development sample [75.0 mL] (18) | | X | | | | | | | | |
| VACCINATION (20) | X | | | | | | | | | |
| Check for AEs following vaccination | X (21) | | | | | | | | | |
| Symptom-driven physical exam (22) | | X | X | X | X | X | X | X | X | X |
| Inspection of injection site of previous vaccinations | | X | | | | | | | | X (25) |
| Explain eDiary (24) | X | | | | | | | | | |
| Review eDiary | | X | | | | | | | | X (26) |
| Check eDiary for SAEs/ AESIs | X | X | X | X | X | Χ | X | X | X | X |
| Scripted Safety Assessment | X | X | X | X | X | X | X | X | X | X |
| AE/ SAE/ AESI Assessment (27) | X | X | X | X | X | X | X | X | X | X |
| Blood Volume [mL] | 0.0 | 12.0 (33);<br>87.0 (34) | 12.0 | 12.0 | 17.0 | 12.0 | 17.0 | 12.0 | 17.0 | 5.0 |

<sup>(1)</sup> Re-screening of subjects is allowed once. Assessments, which have been performed during the first screening visit, remain valid for 14 days. In case re-screening occurs outside this time frame, already performed measures have to be repeated.

Adapted from:
STAT03\_A Statistical Analysis Plan
Confidential and intellectual property of \_\_\_\_\_. No part of this document or its contents may be duplicated, referenced, published or otherwise disclosed in any form or by any means without prior written consent of \_\_\_\_\_.

At on-site Visits, subjects will be supplied with urine pregnancy test kits to ensure that subjects can test for pregnancy at home in case the COVID-19 pandemic prohibits in-person visits at subsequent scheduled visits (Visit 2, 4, 6, 7 and 8). Pregnancy test handling has to be explained to subjects by trained study site staff during Visit 1.

Visit 1A is a safety follow-up visit to be performed 7 days after the first vaccination (i.e. on Day 8). It is intended to perform Visit 1A remotely via a phone/video call in adult subjects (aged 18-65 years) and preferably as an in-person visit in adolescent subjects (aged 12-17 years) and children (5-11 years). If the COVID-19

- pandemic prohibits in-person visits, Visit 1A may also be conducted remotely via a phone/video call in the younger age cohorts. For details on differences in respective study event procedures during in-person or remote visits, please refer to CSP Section 4.2.1.
- Visit should preferably be conducted as an in-person visit. If an in-person is not feasible due to COVID-19, e.g. travel restrictions, local recommendations, circumstances at the study site's location that prohibit an in-person visit, or if the Principle Investigator believes that the subject's safety and well-being might be jeopardized with an in-person visit at the study site due to COVID-19, the visit should be conducted remotely. In case subject visit has to be performed remotely, a mobile nurse professional will come to the subject's home and take the immunogenicity sample within the specified time window. Review of subject eDiary safety data will be performed by the study site via phone/video call. For details on differences in respective study event procedures during in-person or remote visits, please refer to CSP Section 4.2.4. In order to perform urine pregnancy test at home, subjects will be supplied with additional test kits at the last on-site Visit.
- (5) Visit 5A will be performed in a subset of approximately 150 adult subjects only.
- (6) Every effort should be made to have discontinued subjects complete the early termination visit. If the subject is unwilling to perform an Early Termination (ET) visit, a phone-call should be made to follow-up on Adverse Events and Concomitant Medications/ Vaccinations. Note: If a subject presents at a regular study visit and informs the site that it will discontinue the study after this visit, the study visit will not be performed as an ET visit, but as a regular study visit including all events that are described for the respective study and ET visit.
- (7) Informed consent/assent may be obtained within 10 days before Visit 1. For the Booster Phase, subjects are asked to reconfirm the consent/assent within 14 days before Visit 8B.
- (8) Symptoms noted at Visit 1 (prior to first vaccination) are not considered AEs but will be recorded as medical history.
- (9) Physical examination on the following body systems: general appearance (including assessment of body weight and height), skin, head/ eyes /ears/ nose/ throat, chest, lungs, heart, abdomen, extremities and joints, lymph nodes, and neurological system. An Electrocardiogram (ECG) will be performed at Visit 0 only.
- Vital signs (Systolic and diastolic blood pressure and pulse rate while seated and at rest) to be measured prior to vaccination and in addition prior to discharge in case subject reports any complaints.
- (11) To be performed prior to vaccination.
- The results of negative Human Immunodeficiency Virus (HIV) tests that were performed up to 4 weeks before Visit 0 are acceptable (blood: HIV test 3.0 mL). Positive HIV test obtained by ELISA will have to be confirmed by a second method (e.g. Western Blot or Polymerase Chain Reaction (PCR)). HIV tests only in subjects aged ≥ 12 years.
- (13) A commercially available Lyme borreliosis screening test will be performed (blood: 5.0 mL). Serum samples that are tested positive will have to be verified by a confirmatory immunoblot. Test result does not need to be available before randomization and remains valid for 4 weeks.
- (14) In case an ET Visit is performed remotely, the collection of the Lyme borreliosis screening sample will be omitted.
- Female subjects aged ≥12 years and woman of childbearing potential. A woman is considered of childbearing potential if fertile and until becoming post-menopausal unless permanently sterile. A woman that is considered of non-childbearing potential must be e.g. surgically sterilized for at least 3 months prior to Visit 1 (e.g. by hysterectomy, bilateral salpingectomy, bilateral oophorectomy, transcervical sterilization), or postmenopausal for at least one year prior to Visit 1. For serum pregnancy test: tests that were performed in study laboratory within visit window and where results are available at study visit are acceptable. Testing will only be performed in the 5 to 11 age cohort in female subjects after onset of menarche.
- (16) At vaccination visits, all samples have to be obtained before vaccination. Pregnancy results must be available before vaccination.
- (17) Blood will be collected for immunogenicity testing by an IgG binding assay and for supportive functional antibody testing by collected for immunogenicity testing by an IgG binding assay and for supportive functional antibody testing by
- (18) Assay development sera will be collected in adult subjects (age cohort 18 to 65 years) only and will be used for further development of clinical assays.
- (19) To be performed by study staff otherwise not involved with study conduct to keep the study observer-blinded (i.e. un-blinded study staff)
- Preparation of vaccination must be done by designated unblinded staff members (4.2.12) only. Administration of the vaccine can be performed by blinded OR unblinded staff. Vaccination with the assigned treatment has to be administered into the deltoid of the non-dominant arm. Subjects should be observed for at least 30 minutes for treatment of any immediate reactions.
- (21) If subject has any complaints after vaccination, a symptom-driven physical examination will be performed by the investigator prior to discharge.
- Except for Visit 1: Body systems for which the subject reports any symptoms should be evaluated and relevant abnormal findings documented as AEs. At vaccination days the symptom-driven physical exam is to be performed before administration of the vaccination.

Adapted from: STAT03\_A Statistical Analysis Plan Version 6.0, Effective Date 16-Feb-2018 Confidential and intellectual property of

without prior written consent of

- (23) At in-person visits for subjects aged 5-17 years.
- At Visit 1, the subjects will be provided with thermometer and measuring tapes. The subjects will assess solicited local and systemic AEs themselves over a period of seven consecutive days after each vaccination. Subjects/ legal representative(s) will also be instructed to immediately inform the site in case of symptoms suggesting Lyme borreliosis, or any severe solicited AEs or other severe symptoms.
- (25) For Early Termination prior to Visit 6 in Part A or Visit 9 in Part B, the previous injection site should be inspected.
- (26) Subject eDiary entries should be reviewed at the ET Visit if not done at previous visit.
- Unsolicited AEs will be collected within 28 days after each vaccination. SAEs and AESIs will be collected throughout the entire study conduct and documented in the eCRF. Symptoms noted at Visit 1 prior to vaccination are not considered adverse events but will be recorded as medical history.
- (28) In females of non-childbearing potential (before onset of menarche) and male subjects aged <12 years i.e. without serum pregnancy and HIV test
- (29) In females aged <12 years and after onset of menarche i.e. with serum pregnancy test and without HIV test
- (30) In females of non-childbearing potential (surgically sterile or postmenopausal) and in males aged ≥12 years i.e. without serum pregnancy test and with HIV test
- (31) In females aged ≥12 years and of childbearing potential i.e. with serum pregnancy test and HIV test
- (32) A blood draw of in total 75.0 mL will be taken in subjects aged 18-65 years.
- (33) A blood draw of in total 12.0 mL will be taken in subjects from following age cohorts: 5-11 years and 12-17 years.
- (34) A blood draw of in total 87.0 mL (12.0 mL for immunogenicity and 75.0 mL for assay development) will be taken in subjects from age cohort 18-65 years.
- (35) Visit 8B should preferably be performed on the same day as Visit 8.
- (36) If the subject is unwilling to perform an ET visit, a phone call should be made to follow-up on Adverse Events and Concomitant Medications/Vaccinations.
- (37) Only to be performed if V8B is performed more than 14 days after V8, otherwise the assessment is already captured at Visit 8.
- (38) Test results do not need to be available before vaccination.

#### 2. GENERAL CONSIDERATIONS

#### 2.1 Conduct of Analysis

The following analyses are planned:

- Analysis 1 will include all safety and available ELISA immunogenicity data from selected time points from Part A up to Day 208/ Month 7 including the primary endpoint.
  - o Analysis 1.1: Cohort 1, aged 18-65 years
  - o Analysis 1.2: Cohort 2, aged 12-17 years
  - o Analysis 1.3: Cohort 3, aged 5-11 years

Every age cohort can be analyzed separately or might be pooled with age cohorts of previous analyses as soon as data from each cohort is available.

Pooled data from all three cohorts concludes Analysis 1;

- Analysis 2 will include all safety data and available ELISA communication immunogenicity data of Part A up to Month 12 (i.e., 6 months after the third immunization) and will be performed once all subjects have completed Visit 7;
- Analysis 3 will be performed once all subjects have completed Visit 9 (Month 19):
  - Analysis 3.1 will include all safety data and available ELISA COMMITTEE immunogenicity data of Part
     A up to Month 18;
  - Analysis 3.2 will include all safety data and available ELISA communication immunogenicity data from Part B up to Month 19.

Separate statistical analysis outputs will be produced for Analysis 3.1 and Analysis 3.2.

- Analysis 4 will include all safety and ELISA communogenicity data of Part B up to Month 26. The analysis will be performed once all subjects have completed Visit 11;
- Analysis 5 will include all safety and ELISA immunogenicity data of Part B up to Month 30. The analysis will be performed once all subjects have completed Visit 12;
- Analysis 6 will include all safety and ELISA immunogenicity data of Part B up to Month 42. The analysis will be performed once all subjects have completed Visit 14;
- Analysis 7 will include all safety and ELISA immunogenicity data of Part B up to Month 54. The analysis will
  be performed after the last subjects completed the last study visit (Visit 16).

In case analyses fall close in timing, they may be merged.

#### 2.2 Statistical Software and Quality Control

All statistical analyses will be performed using SAS® version 9.3 or higher. Tables, figures and data listings (TLFs) are generated in Microsoft® Word® as well as PDF® format.

Quality control of SAS® programs will include a review of the whole process of result generation:

- Review of all analysis SAS® programs;
- Review of SAS® log for errors, warnings and other notes that could indicate mistakes in the programs;

Adapted from:
STAT03\_A Statistical Analysis Plan

Review of all tables, listings and figures for completeness and correctness.

As additional quality control measure, independent re-programming will be performed as described in Standard Operating Procedure (SOP) SASO4.

#### 2.3 Applicable Standard Operating Procedures

The applicable Standard Operating Procedures (SOPs) of CO for this study are:

STAT03 Statistical Analysis Plan

STAT04 Interim Analysis

STAT05 Randomization and Unblinding

STAT06 Data Review Meeting

STAT07 Report Writing

SAS01 SAS General Principles

SASO4 Handling of Statistical Analyses

SAS06 CDISC- ADaM

SAS07 CDISC - Quality Control

#### 2.4 Randomization and Blinding

Subjects are allocated to study groups via the randomization module of the EDC system. In the Main Study Phase subjects are randomized 1:1:1 to the three study groups, randomization is stratified by age in a 2:1:1 (adults: 18-65 years; adolescents: 12-17; children: 5-11 years) ratio. Date and time of enrollment are defined as the time point at which the subject is randomized.

The study is an observer-blinded study, which is conducted in a blinded manner for the study investigators, the sponsor including laboratory personnel, and the subjects. An overview of persons who will be unblinded and blinded is provided below:

#### **Unblinded:**

- Designated study site staff who randomize subjects to study groups and are concerned with Investigational Medicinal Product (IMP) handling (i.e. perform preparation and maintain drug dispensing log). These unblinded study staff members will not conduct any other study procedures;
- Clinical Research Associates (CRAs) responsible for monitoring of IMP handling and related data for verifying drug accountability during the study and performing overall drug accountability;
- Dedicated statistical team at the Clinical Research Organization (CRO) performing statistical analyses for generation of safety data tables for the Data Safety Monitoring Board (DSMB) and (Internal Review Committee (IRC);
- DSMB members:
- IRC members.

#### Blinded:

- Study participants and legal representative(s);
- Investigators and other study staff involved in general study conduct and safety assessments;

- All other CRAs (responsible for monitoring study data apart from IMP handling/drug accountability);
- All other sponsor/ collaboration partner and CRO staff including laboratory personnel at the sponsor's labs for immunogenicity assessments.

#### Unblinding during the study:

The study sponsor/ collaboration partner and study statisticians will be unblinded at the time of the primary endpoint analysis, i.e. Day 208 analysis, in each age cohort (i.e., Analysis 1.1, Analysis 1.2 and Analysis 1.3) after the respective database snapshot has been performed. All other study personnel including the investigators and other study staff involved in general study conduct and safety assessments as well as laboratory personnel who are performing analytical assays will remain blinded until study end.

#### 2.5 Descriptive Analyses

Descriptive analyses of continuous variables (summary statistics) will be described with the number of non-missing observations, arithmetic mean, standard deviation (±SD), median, quartiles (Q1 and Q3) and range (minimum and maximum).

Descriptive analyses of continuous immunogenicity variables (i.e. tables for the GMT and GMFR) will be described with the number of non-missing observations, geometric mean, confidence intervals for the geometric mean, standard deviation of logarithmic values, median, quartiles (Q1 and Q3) and range (minimum and maximum). Categorical variables (frequency statistics) will be described with the number of non-missing observations and percentages (%). Percentages will be calculated on the total number of non-missing observations, if not stated otherwise.

#### 2.6 Center and Country Effect and Stratification

No country effect will be considered since all centers are located in the United States. The center effect will be taken into account and estimated by adding study site in ANOVA models (sensitivity analyses). Also other covariates will be used as described in Section 5.3.

Furthermore, selected tables will be presented by stratification factor age cohort. If not stated otherwise, the stratification will be implemented by showing the overall data in a first section followed by separate sections for each age cohort separately starting with the oldest age cohort. A separate column in the List of TLFs (Section 7) defines which tables are stratified by age cohort.

#### 2.7 Handling Missing Data

Generally, missing values of immunogenicity variables will not be imputed, and the analyses will be limited to observed values. For missing data in AE evaluation (i.e. missing information if serious, medication taken, severity and causality) a worst case approach will be applied. In case of missing assignment to solicited or unsolicited, this AE will be neither counted in tables for solicited AEs nor in tables for unsolicited AEs but in tables for all AEs. For more details see Section 6.1.3.

Adapted from: STATO3\_A Statistical Analysis Plan Version 6.0, Effective Date 16-Feb-2018 

#### 2.8 Protocol Deviations

In general, Data Review Meetings (DRM) will be conducted on all available data to review protocol deviations, to discuss specific unforeseeable data issues, and to allocate the subjects to the analysis sets. In particular, the respective Per-Protocol Analysis Sets and the Booster Per-Protocol Analysis Sets will be defined in the DRMs. In case analyses fall close in timing, DRMs may be merged. DRMs will be conducted at least prior Analyses 1.1, 1.2 and 1.3 in Part A to define the Per-Protocol Analysis Set and prior Analysis 3.2 to define the Booster Per-Protocol Analysis Set which will be used for the remaining study part. Further DRMs might be conducted prior the respective database snapshots or database closure. Protocol deviations will be classified as "not relevant" or "relevant" deviations on a case by case decision, based on the potential impact on the immunogenicity analysis. Protocol deviations identified by the monitor will be classified as "major" or "minor" by the CRA prior the meetings.

Associated decisions of the DRMs will be documented and approved in the Data Review Meeting Report.

Protocol violations classified as "relevant" during the DRMs and / or classified as "major" by CRA will be described in the CSR (Clinical Study Report).

#### 2.8.1 Part A: Main Study Phase

"Relevant" protocol violations that lead to exclusion from the Per-Protocol Analysis Set in the Main Study Phase (see Section 0) will include the following but are not limited to:

- Subjects with less than three primary vaccinations (Day 1, 57 and 180);
- Subjects who received the wrong IMP;
- Subjects who fulfilled exclusion criteria 2, 8, 9, 13;
- Subjects with substantial time window violations on vaccination visits (Visits 3 and 5)
  - o Target Date of Visit 3 (Day 57) +/-10 days
  - Target Date of Visit 5 (Day 180) +14/-28 days;
- Subjects with other deviations that may affect immune response.

#### 2.8.2 Part B: Booster Phase

"Relevant" protocol violations that lead to exclusion from the Booster Per-Protocol Analysis Set (see Section 2.10.6) will include the following but are not limited to:

- Subjects enrolled despite exclusion from the PPAS of the Main Study Phase;
- Subjects who received the wrong booster IMP;
- Subjects who fulfilled the Booster Phase exclusion criteria 5 and 8;
- Subjects with other deviations that may affect immune response.

#### 2.9 Exclusion of Time Points in the Per-Protocol Analysis

In the Per-Protocol Analysis immunogenicity samples that are outside the predefined time windows described below will be excluded at the respective visit (exclusion of subjects from the Per-Protocol Analysis Set is described in Section 2.8):

Adapted from:  STATO3\_A Statistical Analysis Plan



In the Booster Per-Protocol Analysis immunogenicity samples that are outside the predefined time windows described below will be excluded at the respective visit (exclusion of subjects from the Booster Per-Protocol Analysis Set is described in Section 2.8):

| | Window Per-Pr | Comments | |
|---|---|---|---|
| | Start date | End date | |
| Visit 9 | Visit 8B plus 28 days minus 14days | Visit 8B plus 28 days plus 14days | |
| Visit 10 | Visit 9 plus 4 months minus 28 days | Visit 9 plus 4 months plus 28 days | 4 months = 120 days |
| Visit 11 | Visit 10 plus 3 months minus 28 days | Visit 10 plus 3 months plus 28 days | 3 months = 90 days |
| Visit 12 | Visit 11 plus 4 months minus 36 days | Visit 11 plus 4 months plus 36 days | 4 months = 120 days |
| Visit 13 | Visit 12 plus 6 months minus 36 days | Visit 12 plus 6 months plus 36 days | 6 months = 180 days |
| Visit 14 | Visit 13 plus 6 months minus 36 days | Visit 13 plus 6 months plus 36 days | 6 months = 180 days |
| Visit 15 | Visit 14 plus 6 months minus 36 days | Visit 14 plus 6 months plus 36 days | 6 months = 180 days |
| Visit 16 | Visit 15 plus 6 months minus 36 days | Visit 15 plus 6 months plus 36 days | 6 months = 180 days |

#### 2.10 Analysis Populations

#### 2.10.1 Safety Analysis Set (SAS)

The Safety Analysis Set (SAS) includes all subjects who entered into the study and received at least one vaccination. The SAS will be used for all baseline, safety and tolerability analyses including demographic data, local/systemic tolerability, laboratory data, (S)AEs and AESIs. All analyses based on the SAS will be carried out using the actual treatment received. Details for the derivation of the actual treatment are described in Section 2.12.

#### 2.10.2 Full Analysis Set (FAS)

The Full Analysis Set (FAS) is defined to include all subjects enrolled who received at least one vaccination. Subjects will be analyzed according to the study group they had been allocated to, rather than by the actual treatment they received. If the SAS and FAS Population are identical (i.e. no mistreated) the analysis will be performed for the SAS and the FAS together, labeled with "Safety / Full Analysis Set".

#### 2.10.3 Per-Protocol Analysis Set (PPAS)

The Per-Protocol Analysis Set (PPAS) consists of the FAS population excluding subjects that meet one of the exclusion criteria described in Section 2.8.1). For immunogenicity analysis, the PPAS will be the primary analysis population. The PPAS will be defined for each age cohort in a BDRM prior the respective analysis (i.e. Analysis 1, Analysis 2 and Analysis 3).

#### 2.10.4 Booster Safety Analysis Set (BSAS)

All safety analyses of Part B will be based on the Booster Safety Analysis Set (BSAS), which is defined as all subjects enrolled in Part B who received the booster vaccination. The BSAS will be used for all baseline, safety and tolerability analyses including demographic data, local/systemic tolerability, laboratory data and (S)AEs and AESIs. All analyses based on the BSAS will be carried out using the actual treatment received. Details for the derivation of the actual treatment are described in Section 2.12

#### 2.10.5 Booster Full Analysis Set (BFAS)

The Booster Full Analysis Set (BFAS) is defined as all subjects who received the booster vaccination. Subjects will be analyzed according to the study group they had been allocated to, rather than by the actual treatment they received. If the BSAS and BFAS Population are identical (i.e. no mistreated) the analysis will be performed for the BSAS and the BFAS together, labeled with "Booster Safety / Booster Full Analysis Set".

#### 2.10.6 Booster Per-Protocol Analysis Set (BPPAS)

The Booster Per-Protocol Analysis Set (BPPAS) consists of the BFAS excluding subjects that meet one of the exclusion criteria described in Section 2.8.2. For booster immunogenicity analysis, the BPPAS will be the primary analysis population. The BPPAS will be defined in a BDRM prior the respective Analysis 3.

### 2.11 Subject Data Listings

All vaccinated subjects will be included in the listings, if not stated otherwise. Data listings will include the subject number as identifier (and parameter and/or visit if available) and are sorted by subject ID (and parameter and/or visit if available), if not stated otherwise. The planned study groups will be displayed in listings of the Overall Study Information, Baseline Evaluation (see Sections 0 and 4) and in the immunogenicity listings (see Section 5). Additionally, a column indicating if a subject is in the PPAS is shown in all immunogenicity listings. The actual treatment will be displayed in the safety listings (see section 0).

#### 2.12 Columns in Tables and Derivation of Actual Treatment

 Tables in the overall study information (Section 3), baseline evaluation (Section 4) and unsolicited AEs or other safety results (Section 0) will show one column per study group (i.e. Group 1, Group 2, Group 3), a

Adapted from: STATO3\_A Statistical Analysis Plan Version 6.0, Effective Date 16-Feb-2018 

column for the two pooled VLA15 study groups pooled together with subjects receiving VLA15 at least once but that cannot be assigned to Group 1 or Group 2 and a column showing all vaccinated subjects<sup>2</sup>.

- Tables defined for immunogenicity analysis (Section 5) will show one column for each study group as randomized.
- Tables defined for safety analysis (Section 0) will be presented by following columns:
  - Tables showing Adverse Events after any vaccination will be presented by columns Group 1, Group 2, Group 3, a column for the two VLA15 study groups pooled including subjects that received VLA15 at least once and but cannot be assigned to one of the existing study groups (label "Received any vaccination") and a column for all subjects pooled.

Columns Group 1, Group 2 and Group 3 include

- All subjects that were randomized to the respective study group and received no wrong IMP at any vaccination;
- All subjects that were randomized to a study group but erroneously received the vaccination schedule of another study group. E.g. If a subject was randomized to Group 2 but erroneously received VLA15 instead of placebo at the second vaccination and all other vaccinations were performed as randomized, the subject fulfill the vaccination schedule of Group 1 and is analyzed in Group 1.

Column "Received any VLA15" includes

- o All subjects with actual study treatment of Group 1 and Group 2 as described above;
- All subjects that were mistreated and cannot be allocated to any existing study group as described above, i.e. subjects randomized to Group 2 but that received Placebo instead of VLA15 at the first vaccination and the remaining vaccinations as randomized and thus, cannot be allocated to the vaccination schedules of Group 1, Group 2 or Group 3 and will be analyzed in column "Received any VLA15:
- Adverse Events by vaccination period will be presented by separate tables for each vaccination presented by the columns "VLA15" and "Placebo". Subjects will be allocated to those columns based on the actual treatment they received at the respective vaccination;
- Subjects in Groups 1 and 2 that missed a VLA15 vaccination will only be shown in columns "any VLA15" and "all subjects". Subjects in Group 1 that only missed second vaccination will be shown in column for Group 2 (and "any VLA15" and "all subjects").

In case of a statistical test an additional column showing the p-value will be displayed.

-

 $<sup>^2</sup>$  Pooled VLA15 group column may also contain subjects that received wrong treatment that could not explicitly be assigned to Group 1 or 2

#### 2.13 Medical Coding

Adverse events, medical history and concomitant procedures will be coded using Medical Dictionary for Regulatory Activities (MedDRA) and concomitant medications and vaccination history will be coded using WHO Drug Reference List and Anatomical Therapeutic Chemical (ATC) Classification System as described in the Coding Guideline. Events reported in the adverse events log will be combined with solicited symptoms from the diary section. Solicited symptoms will be coded as described in Section 6.1.3.2.

#### 2.14 Labelling of Visits

The following labels for visits are used in the analysis:

| Visit | Label | Visit | Label |
|---------|-------------------|----------|-----------|
| Visit 0 | V0 (M0/Screening) | Visit 9 | V9 (M19) |
| Visit 1 | V1 (D1) | Visit 10 | V10 (M23) |
| Visit 2 | V2 (M1/D29) | Visit 11 | V11 (M26) |
| Visit 3 | V3 (M2/D57) | Visit 12 | V12 (M30) |
| Visit 4 | V4 (M3/D85) | Visit 13 | V13 (M36) |
| Visit 5 | V5 (M6/D180) | Visit 14 | V14 (M42) |
| Visit 6 | V6 (M7/D208) | Visit 15 | V15 (M48) |
| Visit 7 | V7 (M12/D365) | Visit 16 | V16 (M54) |
| Visit 8 | V8 (M18/D545) | | |

#### 2.15 Changes in the Conduct of the Study or Planned Analysis

Statistical analyses are performed according to CSP. In case any statistical analysis deviates from SAP, all changes are described and justified in the CSR.

#### 2.16 Effect of COVID-19

The study sponsor continuously monitors and evaluates the development of the COVID-19 pandemic in the area of study sites to determine if any measures need to be implemented to mitigate undue risks to the subjects or in response to local governmental recommendations. Such measures may include, temporarily halting further recruitment, switching in-person visits to phone/video calls, or employing mobile teams to collect serum samples.

In particular, visits should preferably be conducted as in-person visits. Instead of in-person visits, visits can be conducted remotely due to COVID-19 (e.g., phone/video call) for Visits 2, 4, 5A, 6, 7, 8 and early termination visit as described in the CSP. It is tabulated and listed whether visits were performed remotely or in-person. In case subject visit has to be performed remotely, a mobile nurse professional will come to the subject's home and take the immunogenicity sample within the specified time window. Review of subject eDiary safety data will be performed by the study site via phone/video call.

At on-site visits, subjects are supplied with urine pregnancy test kits to ensure that subjects can test for pregnancy at home in case the COVID-19 pandemic prohibits in-person visits at subsequent scheduled visits (Visit 2, 4, 6, 7).

and 8). If the COVID-19 pandemic prohibits in-person visits, Visit 1A may also be conducted remotely via a phone/video call in the younger age cohorts.

COVID-19 vaccinations interfering with the IMP are subject to review in the DRM for possible exclusion from the PP. During the DRM, protocol deviations will be classified as COVID-19-related or not COVID-19-related.

#### OVERALL STUDY INFORMATION

Analyses will be performed for the SAS, FAS and PPAS for Part A and analyses of Part B will be performed on BSAS, BFAS and BPPAS. In case (B)SAS and (B)FAS are identical, Section 2.10.2 for Main Study Phase and Section 2.10.5 for Booster Phase apply.

#### 3.1 Data Points

The following information will be analyzed descriptively and corresponding details on the subject level will be provided in data listings:

- · Subject overview
- Screening failures and reasons
- Randomization
- Violated inclusion/exclusion criteria (will only be listed)
- · Study vaccination details
- Visits details
- Attendance status and early termination details
- · Protocol deviations
- Visits performed remotely

Specifications on tables and listings are provided in the List of TLFs (see Section 7).

#### 3.2 Definitions

- Screening failures will be identified by checking if the "Visit attendance status of subject" is answered with "screening failure" on the eCRF page "End of Study";
- For Analysis 1.1/1.2/1.3 and Analysis 1 the cut-off for early termination data is defined by Day 208/ Month 7;
- For Analysis 2 the cut-off for early termination data is defined by Day 365/ Month 12;
- For Analysis 3.1 the cut-off for early termination data is defined by Month 18 (i.e. includes all available data for Main Study Phase subjects);
- For Analysis 3.2 the cut-off for early termination data is defined by Month 19;
- For Analysis 4 the cut-off for early termination data is defined by Month 26;
- For Analysis 5 the cut-off for early termination data is defined by Month 30;
- For Analysis 6 the cut-off for early termination data is defined by Month 42;
- For Analysis 7 all available early termination data are analyzed;

 Early terminations up to data cut-off will be detected by calculating the last attended scheduled visit for subjects with visit attendance status "early termination" on the End of Study page in the eCRF.

#### 4. BASELINE EVALUATION

Analyses will be performed for the SAS, FAS and PPAS for Part A and analyses of Part B will be performed for BSAS, BFAS and BPPAS. In case (B)SAS and (B)FAS will be identical, Section 2.10.2 for Main Study Phase and Section 2.10.5 for Booster Phase applies.

#### 4.1 Data Points

The following information will be analyzed descriptively and corresponding details on the subject level will be provided in data listings:

- Demographic Information (gender, childbearing potential, age [years], age cohort, race, ethnicity, body height [cm], body weight [kg] and body mass index [kg/m²])
- Physical examination (is only listed)
- ECG
- Vaccination history
- Medical History
- Prior/Concomitant Procedures
- Prior/Concomitant Medication
- HIV (is only listed)

#### 4.2 Definitions

- Baseline analyses is based on data of Visit 0;
- Body height will be analyzed in centimeters (cm). Body height documented in inch (in) will be converted to cm using the following rule: height [cm] = height [in] × 2.54;
- Body weight will be analyzed in kilogram (kg). Body weight documented in pounds (lbs) will be converted to kg using the following rule: weight [kg] = weight [lbs] × 0.45359237;
- The Body Mass Index [kg/m2] will be calculated as (kg/cm2) × 10,000
- Medications / Procedures stopped prior (<) to Day 1 (Visit 1) will be considered prior medications /procedures, all other medications procedures will be considered to be concomitant. Medications / Procedures with a missing or incomplete end date where it cannot clearly be decided if the end date was before or after Day 1 (Visit 1) will be considered concomitant:</p>
- For Analysis 1.1/1.2/1.3 and Analysis 1 the cut-off for medications / procedures data is defined by Day 208/ Month 7;
- For Analysis 2 the cut-off for medications / procedures is defined by Day 365;
- For Analysis 3.1 the cut-off for medications / procedures is defined by Month 18 (i.e. includes all available data for Main Study Phase subjects);

Adapted from:  STATO3\_A Statistical Analysis Plan

- For Analysis 3.2 the cut-off for medications / procedures is defined by Month 19 (i.e. includes all available data from Main Study Phase for Booster subjects);
- For Analysis 4 the cut-off for medications / procedures is defined by Month 26;
- For Analysis 5 the cut-off for medications / procedures is defined by Month 30;
- For Analysis 6 the cut-off for medications / procedures is defined by Month 42;
- For Analysis 7 all available medications / procedures are analyzed:
- Medications/procedures will be considered to have started up to data cut-off if the start date of the medication/procedure is before or on data cut-off (e.g. Day 208/ Month 7 for Analysis 1). In case of an incomplete start date where it cannot clearly be decided if the medication/procedure started up to data cut-off or not, the medication/procedure will be considered to have started up to data cut-off. For derivation of cut-off, the date of the respective Visit is used (e.g. date of Visit 6 for Day 208, date of Visit 7 for Day 365). In case no respective visit was performed, the cut-off is determined as date of Visit 1 plus number of days minus 1 (e.g. date of Visit 1 +207 if no Visit 6 date is available). For distances between visits defined as month, see Section 2.9;
- Medical history not stopped prior (<) to informed consent will be considered ongoing at study entry. Entries with a missing or incomplete stop date where it cannot clearly will be decided if the stop date was before or after informed consent will be considered ongoing at study entry.
- Prior vaccinations erroneously reported in the concomitant medication section of the eCRF instead of the section "Vaccination history" will be excluded from the tables showing prior medications. Those entries will be detected by using the ATC level 2 "Vaccines" and will be added to the summary count in the vaccination history table.

#### 5. IMMUNOGENICITY ANALYSIS

All immunogenicity analyses will be performed on the PPAS and will be repeated for selected analyses on the FAS for Part A. For Part B, all immunogenicity analyses are available for BPPAS and selected analyses will be repeated for the BFAS. Selected TLFs will be repeated for the different age cohorts. Specifications are given in Section 7. The primary immunogenicity analysis will be based on the PPAS for the Main Study Phase and based on the BPPAS for the Booster Phase.

All immunogenicity analyses will contain all available time points, i.e. time points which were already analyzed in previous analyses will be repeated in the current analysis. All immunogenicity time points of Part A will further be repeated in Part B based on the respective booster analysis population, if not stated otherwise.

For the evaluation of immunogenicity, human sera will be analyzed for IgG against each OspA serotype (ST1 to ST6) separately by a quantitative ELISA. ELISA immunogenicity data are available in Part A at Visit 0 and Visit 4 to Visit 8 as well as in Part B for Visits 9 to Visit 16.



#### 5.1 Data Points

#### 5.1.1 Tables and Listings

The following information will be analyzed separately for ELISA collections and for both study parts A and B, if not stated otherwise. Corresponding details on subject level will be provided in data listings.

Summary tables for categorical immunogenicity variables:

- Immunogenicity blood sample availability by time point
- ELISA:
  - Immunogenicity results/serostatus (report concentration/negative;) by OspA specific serotype
     by time point (including baseline serology status)
  - Subjects by OspA specific IgG serostatus by visit
  - o SCRs for OspA specific IgG antibodies by visit
    - each OspA serotype (separate tables for ST1 to ST6)
    - all six OspA serotypes combined
    - ST1 and ST2 combined



Summary tables for continuous immunogenicity variables are provided:

#### • ELISA:

- GMTs for IgG against each OspA specific serotype (ST1 to ST6) by visit (separate table for each OspA serotype).
- GMFRs as compared to Visit 0 for IgG against each OspA serotype by visit (separate tables for each OspA serotype)
- GMFRs as compared to Day 208 for IgG against each OspA serotype by visit (separate tables for each OspA serotype, only applicable for Part B)
- GMFRs as compared to Month 12 for IgG against each OspA serotype by visit (separate tables for each OspA serotype, only applicable for Part B)



 GMFRs as compared to Month 18 for IgG against each OspA serotype by visit (separate tables for each OspA serotype, only applicable for Part B)



#### **Correlation Analysis:**

- ELISA:
  - Correlation analyses for each OspA Specific IgG titer with each other OspA specific IgG titer, respectively, at Day 208 and Month 19 (15 comparisons in total for each time point; pooled VLA15 study groups and for each VLA15 study group separately; IgG ELISA seropositive samples at Screening will be excluded from the correlation analysis)



Inferential analysis will be performed as described in Section 5.3. Details are specified in Section 7.

#### 5.1.2 Figures for ELISA CCI

- ELISA:
  - Bar chart: OspA-specific IgG antibodies (GMT) including 95% confidence intervals for the GMT vs
     OspA specific serotypes by study group for each time point separately (y-axis: GMT; x-axis: OspA specific serotypes per study group)

- Bar chart: OspA-specific IgG antibodies (GMT) including 95% confidence intervals for the GMT by serotype over time for study group 1 and 2 separately (y-axis: GMT; x-axis: serotypes)
- Bar charts: OspA-specific IgG antibodies (GMT) including 95% confidence intervals for the GMT by serotype and age cohort at Day 208 and Month 19 for study groups 1 and 2 separately (y-axis: GMT; x-axis: serotypes)
- Bar charts Seroconversion Rate:
  - Seroconversion Rate by OspA-specific IgG and study group (for each time point separately, y-axis: percentage of subjects, x-axis: OspA STs per study groups)
  - Seroconversion Rate for all OspA-specific IgG serotypes combined over time vs. study group (y axis: percentage of subjects, x axis: visits per study groups; Time points of Part A will not be repeated in Part B)
  - Seroconversion Rate for OspA-specific IgG serotypes ST1 and ST2 combined over time vs.
     study group (y axis: percentage of subjects, x axis: visits per study groups)
- Line charts (y-axis: GMT, x-axis: study days): OspA specific IgG antibodies (GMT) over time vs. study group for each ST1-6 separately
- Line charts (y-axis: GMT, x-axis: study days): OspA specific IgG antibodies (GMT) over time vs.
   serotype for each study group separately
- For each OspA serotype and study group: Reverse cumulative distribution curves for percentage of subjects reaching certain OspA specific IgG titer over time
- For each OspA serotype and study group: Reverse cumulative distribution curves at Day 208 and
   Day 365 for percentage of subjects reaching certain OspA specific IgG titer by age cohort
- Scatter plots representing the correlation between OspA specific IgG antibodies GMTs for each combination of two different OspA specific serotypes for all study groups pooled.

| • | CCI |
|---|-----|
| | _ |
| | _ |



#### 5.2 Derivations and Definitions

• Baseline for immunogenicity ELISA column analysis is defined as Visit 0.

#### 5.2.1 ELISA

- Baseline OspA IgG seropositive/seronegative for ELISA is defined as follows:
  - ELISA samples scored as "negative" or below the quantitation limit of the ELISA (40 U/mL) will be replaced by 20 U/mL;
  - Subjects with screening values below the quantitation limit of the ELISA (40 U/mL) and samples scored as "negative" (i.e. replaced by 20 U/mL) will be considered "baseline OspA IgG seronegative" for each serotype.
  - Subjects with screening values of 40 U/mL and above will be considered "baseline OspA IgG seropositive" for each serotype.
  - Seroconversion for ELISA is defined as:
    - For subjects that are seronegative at screening: a change from seronegative at screening to seropositive (i.e. antibody titer of ≥40 U/mL) at a certain time point.
    - o For subjects that are seropositive at screening: a ≥ 4-fold rise in OspA IgG antibody titer from screening. A subject reaches a 4-fold increase in ELISA if the value at a certain visit after screening is at least 4-times higher than the value at screening. In case of missing values (missing at baseline or current time point), seroconversion will not be calculated.

| CCI |
|-----|



#### 5.3 Statistical Tests

- In general, all statistical tests comparing study groups in the immunogenicity analysis will include all study groups (i.e. Study Group 1, Study Group 2 and Study Group 3).
- ANOVAs with factors study group and age cohort will be performed for the comparison between Study Group
   1, Study Group 2 and Study Group 3 for each OspA ST1 to ST6 respectively. For Interim Analysis A1.1, no
   factor age cohort will be used. The primary immunogenicity analysis of the Main Study Phase is the ANOVA
   for ELISA GMTs at Day 208 in the PPAS.
- This will be done using log10 transformed data and taking the anti-log of the resulting point estimates for the least squares means, least squares means differences and the corresponding 95 % Cls. Tukey's HSD test will be applied for pair-wise comparisons.
- The primary immunogenicity analysis will provide 95% Confidence Intervals for Geometric Mean Titers (GMTs).
- ELISA:
  - ANOVAs will be performed for GMTs as well as GMFRs compared to screening at all available time points.
  - For Part B, ANOVAs will be additionally performed for GMFRs compared to Day 208 and Month 18 at all available time points after Month 18.

- Part A: Sensitivity analyses for GMTs and GMFRs at Day 208 will be performed for ANOVAs with factors study site, study group, age cohort, age cohort\*study group and baseline B.b. s.l serostatus at screening.
- Part B: Sensitivity analyses for GMTs and GMFRs at Month 19 will be performed for ANOVAs with factors study site, study group, age cohort, age cohort\*study group and *B.b.* s.l serostatus at Month 18.
- Summary tables for the OspA specific IgG titer against each OspA serotype and summary tables for the geometric mean fold-rise against each OspA serotype will be amended by an overall test (Kruskal-Wallis).
- SCRs will be compared using Fisher-Freeman-Halton tests, a significant overall test will be amended by pair-wise tests (Fisher's exact test).
- A non-parametric correlation analysis (Spearman) between OspA IgG antibodies GMTs for each combination of two different OspA specific IgG types will be performed for Day 208 and Month 19, Study Group 1 and Group 2 separately as well as for all VLA15 study groups together (pooled analysis).

| <del></del> |
|-------------|

#### SAFETY ANALYSIS

Safety Analysis will be performed on SAS for Part A and based on BSAS for Part B. Data from early termination and unscheduled visits will be listed only, if not states otherwise.

#### 6.1 Adverse Events

#### 6.1.1 Documentation of Adverse Events

In general, there are four sources in the eCRF for AEs: Assessment after vaccination, AE Log, eDiary and Reviewed eDiary.

- The subjects should be kept under medical supervision for at least 30 min after vaccination. Any findings on solicited AEs have to be documented in eCRF section "Assessment after vaccination".
- All subjects record solicited AEs for the first seven days after each vaccination (starting on the day of vaccination) in eCRF Section "eDiaries".
- The eDiary entries will be reviewed by a clinician together with the subject and the investigator performs an assessment by vaccination period (source "Reviewed eDiary" in eCRF). Severity categories of investigator's assessment are not necessarily identical to the categories provided in the eDiary.
- A) Unsolicited AEs will be reported in the eCRF section "AE Log" up to 28 days after each vaccination. Thereafter, only SAEs and AESIs will be documented in the eCRF.
  - B) Serious and/ or medically attended or solicited systemic Grade 3/4 reactions will also be documented in the eCRF "AE Log". For solicited local and systemic AEs persisting beyond Day 6 after vaccination, the stop date will also be documented in the "AE Log".

#### 6.1.2 Data Points

The following information will be analyzed descriptively and corresponding details on the subject level will be provided in data listings:

#### General (solicited and unsolicited AEs):

- Adverse Events Overview (solicited and unsolicited, including stratification by age cohort)
- Adverse Events Overview (solicited and unsolicited, including stratification by age cohort) by vaccination period
- Serious and related Serious Adverse Events (solicited and unsolicited) by SOC and PT
- Medically attended and related medically attended Adverse Events (solicited and unsolicited) by SOC and PT
- Adverse Events (solicited and unsolicited) leading to withdrawal from further vaccination by SOC and PT (Only applicable for Analysis 1 and it's sub-analyses)
- Adverse Events (solicited and unsolicited) leading to withdrawal from study by SOC and PT
- Non-Serious solicited and / or unsolicited AE by SOC and PT for PTs with Frequency >5 % in any study group
- Non-Serious solicited and / or unsolicited AE by SOC and PT for PTs with Frequency >10 % in any study group

Adapted from: STAT03\_A Statistical Analysis Plan Version 6.0, Effective Date 16-Feb-2018 
# Solicited AE Tables (eCRF Section "Subject Diary" combined with "Reviewed eDiary" and "Assessment after vaccination")

- The following tables will be provided after any vaccination
  - Solicited Adverse Events (by symptom, by maximum severity)
  - Severe solicited Adverse Events (by symptom)
  - Solicited local Adverse Events (by symptom, by maximum severity, separately for symptoms meeting FDA grading scale only)
  - Solicited systemic Adverse Events (by symptom, by maximum severity)
- The following tables will be provided by vaccination period
  - Solicited Adverse Events (by symptom, by maximum severity)
  - Severe solicited Adverse Events (by symptom)
  - Solicited local Adverse Events (by symptom, by maximum severity, separately for symptoms meeting FDA grading scale only)
  - Solicited systemic Adverse Events (by symptom, by maximum severity, )
- The following tables will be provided by diary day
  - Solicited Adverse Events (overall and by symptom)
  - o Mean duration (in days) of solicited Adverse Events by symptom
  - o Greatest single diameter (in cm) for present Erythema, Swelling and Induration
  - Body Temperature (in °C) for case of fever
- The following figures will be provided:
  - Bar chart: The number and percentage of subjects with solicited local Adverse Events by symptom and overall, by study group and grade for the diary period after each vaccination and for the whole treatment period.
  - Bar chart: The number and percentage of subjects with solicited local Adverse Events reaching
     FDA Grading Scale by symptom and overall, by study group and grade for the diary period after each vaccination and for the whole treatment period
  - Bar chart: The number and percentage of subjects with solicited systemic Adverse Events by symptom and overall, by study group and grade for the diary period after each vaccination and for the whole treatment period.

# Unsolicited AE Tables (eCRF Section "Adverse Event Log) for specific types of AEs (e.g. any unsolicited AE, any unsolicited SAE)

- Unsolicited Adverse Events by SOC and PT (overall and additionally for types: related, related serious, severe, related severe and AESI)
- Unsolicited Adverse Event by Maximum Severity (overall and additionally for types medically attended AE and AESI)
- Unsolicited Adverse Event by Causality (overall and additionally for types medically attended and AESI)
- Adverse Events of Special Interest by SOC and PT

Adapted from: STATO3\_A Statistical Analysis Plan Version 6.0, Effective Date 16-Feb-2018 Confidence intervals and statistical tests will be performed as described in Section 6.1.3. Details are specified in Section 7.

#### 6.1.3 Derivations and Definitions

## 6.1.3.1 General Principles for Analysis of Adverse Event

- In general the unsolicited AEs will be taken from the eCRF section "AE-log" and the solicited AEs will be derived from the eCRF sections "Assessment after Vaccination", "eDiary" and "Review of eDiary". For summaries and listings of solicited and unsolicited medically attended AEs and/or serious AEs, the eCRF section "AE-log" will be used as basis rather than taking those AEs from the diary. More details of the derivation of the solicited AEs are given in section 6.1.3.2.
- Tables showing "severe" events will include events with grade 3 or 4 or missing grade.
- For tables by maximum severity and worst causality, subjects will be only counted once in highest grading category and events are counted in each reported grading category.
- Percentages in tables that do not present data by time periods will be based on N (study group totals), if not stated otherwise.
- For Analysis 1.1/1.2.2/1.3 and Analysis 1 the cut-off for AEs is defined by Day 208
- For Analysis 2 the cut-off for AEs is defined by Day 365
- For Analysis 3.1 the cut-off for AEs is defined by Month 18 (i.e. includes all available data for Main Study Phase subjects)
- For Analysis 3.2 the cut-off for AEs is defined by Month 19
- For Analysis 4 the cut-off for AEs is defined by Month 26
- For Analysis 5 the cut-off for AEs is defined by Month 30
- For Analysis 6 the cut-off for AEs is defined by Month 42
- For Analysis 7 all available AEs are analyzed (up to Month 54)
- AEs in the "AE log" will be considered to have started up to cut-off (e.g. Day 208) if the start date of the AE is before or on study day of the cut-off (e.g. date of Visit 6 (Day 208)). In case of an incomplete start date where it cannot clearly be decided if the AE started up to cut-off day or not, the AE will be considered to have started up to the cut-off. For derivation of cut-off, the date of the respective Visit is used (e.g. date of Visit 6 for Day 208, date of Visit 7 for Day 365). In case no respective visit was performed, the cut-off is determined as date of Visit 1 plus number of days minus 1 (e.g. date of Visit 1 +207 if no Visit 6 date is available). For distances between visits defined as month, see Section 2.9;
- For the analysis of non-serious solicited and unsolicited AE the following applies: Solicited AEs (eCRF section "Subject Diary" considering "Reviewed eDiary" and "Assessment after Vaccination") will be considered as non-serious AEs if "no" is ticked for question "Symptom fulfilling any SAE criteria" and unsolicited AEs (eCRF section "Adverse Event log") will be considered as non-serious if "Serious" is ticked with "no". Adverse Events will be only included for this analysis if their occurrence by PT in at least one study group in the Safety Population is 5 % or over 10 %, respectively.

Adapted from:  STATO3\_A Statistical Analysis Plan

#### 6.1.3.2 Principles for Solicited Adverse Events

- In general, for tables summarizing solicited AEs, only the Subject Diary considering the Investigator's review and the "Assessment after vaccination" will be used.
- AE tables presented after any or after each vaccination will be based on the eCRF section "reviewed eDiary" and "Assessment after vaccination". Only available events in these eCRF section will be considered. If a subject has documented its symptoms in the eDiary section but no corresponding event in the eCRF section "reviewed eDiary" is available, the event will not be included.
- The overall maximum severity for each subject is derived using the sources "reviewed eDiary" and "Assessment after Vaccination":
  - The overall maximum severity by subject and each symptom is defined as the maximum of the documented Investigator assessment in the eCRF section "reviewed eDiary" and the severity entered in the eCRF section "Assessment after Vaccination". In case investigator assessment in the eCRF section "reviewed Diary" is not available, the maximum severity which was automatically populated from eCRF source "eDiary" into the eCRF Section "reviewed eDiary" will be used.
  - For symptoms Erythema/Redness and Fever, no automatically populated maximum severity from eCRF source "eDiary" is available. This will be calculated as described in the CSP up to Grade 3:

Table 4: Grading of Erythema and Fever according to CSP (Table 8)

| Symptom | Age | Grade 1<br>Mild | Grade 2<br>Moderate | Grade 3<br>Severe |
|---|---|---|---|---|
| Injection Site<br>Erythema or<br>Redness <sup>1</sup> | 5-11<br>years <sup>(B)</sup> | 1.0 - ≤ 2.5 cm (0.39-<br>0,98 inch) in<br>diameter | > 2.5 - 5.0 cm (2) in<br>diameter with < 50%<br>surface area of the<br>extremity segment<br>involved (e.g., upper<br>arm or thigh) | > 5 cm (2) OR ≥ 50% surface<br>area of the extremity<br>segment involved (e.g.,<br>upper arm or thigh) OR<br>Ulceration OR Secondary<br>infection OR Phlebitis OR<br>Sterile abscess OR Drainage |
| | 12-65 | 2.5-5 cm | 5.1-10 cm | >10 cm |
| | years <sup>(A)</sup> | (0.98-1.96 inch) | 1.97-3.94 inch | >3.94 inch |
| Fever <sup>(4)</sup> | 5-65 | 38.0-38.4/ | 38.5-38.9/ | 39.0-40/ |
| (°C)/(°F) | years <sup>(A)</sup> | 100.4-101.1 | 101.2-102.0 | 102.1-104 |

In case of no available severity investigator assessment in eCRF section "Reviewed eDiary", the grading will be based on the subject's grading in source "eDiary" as described above. For symptom Erythema/Redness for subject aged 5-11 years, this will be done by considering the diameter only but not taking aspects "with < 50% surface area of the extremity segment involved" for Grade 2 and "OR  $\ge 50\%$  surface area of the extremity segment involved (e.g., upper arm or thigh) OR Ulceration OR Secondary infection OR Phlebitis OR Sterile abscess OR Drainage" for Grade 3 in account because this information is not available in the eDiary source.

Adapted from: STATO3\_A Statistical Analysis Plan Version 6.0, Effective Date 16-Feb-2018 

- The presence of symptoms for tables presented by diary day will be based on the eCRF section "reviewed Diary" considering presence information which was populated by the eCRF from Section "eDiary" into "reviewed eDiary". In case the information about the presence of a symptom was revised by the Investigator, the Investigator information will be analyzed (section "reviewed Diary").
- Solicited AEs comprise reactions at the injection site or systemic reactions that are typical for vaccinations.
  - Solicited local AEs are the following injection site reactions: pain, tenderness, induration/ hardening, swelling and erythema/ redness.
  - Solicited systemic AEs are: headache, myalgia (muscle pain), arthralgia (joint pain), fever (oral body temperature), nausea, vomiting and fatigue.
- Solicited AEs are per definition regarded as related to IMP.
- For tables that summarize solicited AEs over several diary days / diary periods, the worst severity of all diary days / diary periods will be taken as the events severity.
- Percentages in tables for solicited AEs by diary period /diary day will be based on the number of subjects
  with available information (diary completed or symptom present on at least one day). In particular, if a
  symptom was not assessed at a certain diary day and the symptom is reported as not present on the other
  days, the subject is not included in the table of the respective symptom and diary period.
- For the derivation of the duration of solicited Adverse Events by symptom and vaccination period the difference of the first occurrence and the last occurrence of the concerning event in the respective vaccination period will be taken, no matter if the event is continuous or not. Therefore, also the end-date if ongoing after day 6 will be considered. If the AE was ongoing after day 6 but has a missing or incomplete end date, the date of last attended visit will be used as end date.
- For swelling, redness and induration, the maximum diameter per diary period in cm will be derived as taking the maximum of all diameters reported in that period for that symptom and converting via [cm] = [in] × 2.54.
- The maximum body temperature per diary period for present symptom fever will be derived as taking the
  maximum temperature of all temperatures reported in that period and converting via [°C] = ([°F] 32) ×
  5/9.
- Adverse Events from the Subject Diary will be coded according to the table below:

Adapted from: STATO3\_A Statistical Analysis Plan Version 6.0, Effective Date 16-Feb-2018

| Event | SOC name | SOC code | PT name | PT code |
|---|---|---|---|---|
| Fatigue | General disorders and | 10018065 | Fatigue | 10016256 |
| | administration site conditions | | | |
| Fever | General disorders and | 10018065 | Pyrexia | 10037660 |
| | administration site conditions | | | |
| Headache | Nervous system disorders | 10029205 | Headache | 10019211 |
| Nausea | Gastrointestinal disorders | 10017947 | Nausea | 10028813 |
| Vomiting | Gastrointestinal disorders | 10017947 | Vomiting | 10047700 |
| Erythema/Redness | General disorders and | 10018065 | Injection site | 10022061 |
| | administration site conditions | | erythema | |
| Induration/Hardening | General disorders and | 10018065 | Injection site | 10022075 |
| | administration site conditions | | induration | |
| Muscle pain | Musculoskeletal and | 10028395 | Myalgia | 10028411 |
| | connective tissue disorders | | | |
| Pain (pain without | General disorders and | 10018065 | Injection site | 10022086 |
| touching) | administration site conditions | | pain | |
| Swelling | General disorders and | 10018065 | Injection site | 10053425 |
| | administration site conditions | | swelling | |
| Joint pain | Musculoskeletal and | 10028395 | Arthralgia | 10003239 |
| | connective tissue disorders | | | |
| Tenderness (pain | General disorders and | 10018065 | Injection site | 10022086 |
| upon touching) | administration site conditions | | pain | |

#### 6.1.3.3 Principles for Unsolicited Adverse Events

- AEs in the AE log will be coded using the MedDRA version that is current at time point of the respective data snapshots and database closure. The version used will be indicated in the respective tables and listings and is documented in the CSR.
- Adverse events in the AE log will be considered related if the causality to IMP is reported as "probable" or "possible" (or missing causality)
- An AE in the AE-log will be considered as "leading to withdrawal from further vaccination" if for "action taken on IMP", "second dose not administered" or "third dose not administered" is ticked.
- An AE in the AE-log will be considered as "leading to withdrawal from study" if in section "other action taken" the question "Withdrawn from study", is answered with "yes".
- Percentages in tables for unsolicited events or all events (solicited and unsolicited) over the whole study will be based on N (study group totals).

Adapted from: STAT03\_A Statistical Analysis Plan Version 6.0, Effective Date 16-Feb-2018

- For presentation of unsolicited AEs by vaccination period, a vaccination period is defined as the period 28 days after each vaccination.
  - 1st vaccination period: AE with start date/time at or after date/time of 1st vaccination and within 28 days of 1st vaccination. If no AE start time is given, the AE will be included if the start date is at or after the date of 1st vaccination and within 28 days of 1st vaccination.
  - Vaccination periods for 2<sup>nd</sup>, 3<sup>rd</sup> and booster vaccination period are defined analogously
  - If a subject did not receive a certain vaccination, the respective vaccination period will not be defined.
  - o In case of incomplete start dates where it cannot be clearly decided to which vaccination period the AE can be assigned, the AE will be assigned to the last received vaccination.

### 6.1.4 Confidence Intervals and Statistical Tests

95 % confidence intervals according to Altman will generally be provided for all AE rates. Differences between the three study groups will be assessed for significance using Fisher's exact (Fisher-Freeman-Halton) test, whereby a significant overall test will be amended by pair-wise tests.

It is stated in detail in Section 7.1.4 for which tables such comparisons are made.

## 6.2 Lyme Borreliosis Screening

# 6.2.1 Data Points

Borrelia burgdorferi s.l. screening tests will be analyzed descriptively at scheduled or early termination visits. All results (i.e. including unscheduled visits, early termination visit and scheduled visits) are listed on subject-level.

- Lyme Borreliosis Screening results by visit (frequency statistics);
- Seroconversion rate of Lyme Borreliosis Screening from Visit 0 to Visit 8/ET (frequency statistics);
- Seroconversion rate of Lyme Borreliosis Screening from Visit 8 to Visit 12/ET (frequency statistics);;
- Seroconversion rate of Lyme Borreliosis Screening from Visit 12 to Visit 14/ET (frequency statistics);
- Seroconversion rate of Lyme Borreliosis Screening from Visit 14 to Visit 16/ET (frequency statistics).

#### 6.2.2 Derivations and Definitions

- In case no result is available at Visit 8 because the subject terminated early, the result from the Early Termination Visit will be considered instead. Same applies for Visit 12, 14 and 16;
- Seroconversion is defined as change from *B.b.* s.l. serostatus "negative" at Visit 0 to *B.b.* s.l. serostatus "positive" at Visit 8/ET for Main Study Phase. Seroconversion rate from Visit 8 to Visit 12, Visit 12 to visit 14 and Visit 14 to Visit 16 will be determined in the same manner. In general, seroconversions will only be determined in case both results (i.e. Visit 0 and Visit 8/ET for Main Study Phase, Visit 8 and Visit 12/ET for Analysis 5, Visit 12 and 14/ET for Analysis as well as Visit 14 and Visit 16/ET for Analysis 7) are available.
- Seroconversion rate will be based on baseline seronegative subjects.

Adapted from: STAT03\_A Statistical Analysis Plan Version 6.0, Effective Date 16-Feb-2018

# 6.3 Other Safety Parameters

The following information will be analyzed descriptively from scheduled visits and corresponding details on the subject level of all visits will be provided in data listings:

- Systolic blood pressure by time point incl. measurements after vaccinations (summary statistics)
- Diastolic blood pressure by time point incl. measurements after vaccinations (summary statistics)
- Pulse rate by time point incl. measurements after vaccinations (summary statistics)
- Oral body temperature by time point (summary statistics)

The following information will only be listed:

- Physical Examination
- Pregnancy Test
- Injection Site Inspection
- Assessment after Vaccination (except solicited Adverse Events documented during post-vaccination assessment, see Section 0)
- Vaccination delay criteria

Adapted from:

STATO3\_A Statistical Analysis Plan


Confidential and intellectual property of \_\_\_\_\_\_. No part of this document or its contents may be duplicated, referenced, published or

otherwise disclosed in any form or by any means without prior written consent of



In general, the numbering consists of the following components in the given order:

| Description | Values |
|---|---|
| CSR Section | 14 = Tables and figures |
| | 16.2 = Listings |
| Analysis number | 1.1 = Analysis 1.1 |
| | 1.2 = Analysis 1.2 |
| | 1.3 = Analysis 1.3 |
| | 1 = Analysis 1 |
| | 2 = Analysis 2 |
| | 3.1 = Analysis 3.1 |
| | 3.2 = Analysis 3.2 |
| | 4 = Analysis 4 |
| | 5 = Analysis 5 |
| | 6 = Analysis 6 |
| | 7 = Analysis 7 |
| Analysis Section | 1 = Overall study information tables / listings |
| | 2 = Baseline evaluation tables / listings |
| | 3 = Immunogenicity analysis tables / listings |
| | 4 = Adverse events tables / listings |
| | 5 = Other safety and B.b. s.l. information tables / listings |
| | 6 = Immunogenicity figures |
| | 7 = Safety figures |
| Analysis Set and label | [Booster] Safety Analysis Set |
| for TLF headers | [Booster] Full Analysis Set |
| | [Booster] Per-Protocol Analysis Set |
| | Note: The analysis set which will be first produced within the statistical output will be |
| | numbered by 1, the number of the further analysis sets continuous depending on the |
| | order of appearance. |
| TLF ID | 1 |
| | 2 |

The population digit is used only in case TLFs are produced for more than one Analysis Set. Further digits can be introduced during the programming of the analysis, if necessary (e.g. introducing sub-continuous numbering in case Listing 16.2.1.1 has to be divided in 16.2.1.1.1 and 16.2.1.1.2).

TLFs showing data up to a certain time point are marked as "[Time Points]". This will be replaced by the following:

Adapted from: STAT03\_A Statistical Analysis Plan Version 6.0, Effective Date 16-Feb-2018

# Part A:

| Analysis | A1.1 | A1.2 | A1.3 | A1 | A2 | A3.1 |
|----------|---------|---------|---------|---------|----------|----------|
| up to | Day 208 | Day 208 | Day 208 | Day 208 | Month 12 | Month 18 |

## Part B:

| Analysis | A3.2 | A4 | A5 | A6 | A7 |
|----------|----------|----------|----------|----------|----------|
| up to | Month 19 | Month 26 | Month 30 | Month 42 | Month 54 |

# 7.1 List of Tables

# 7.1.1 Overall Study Information

| | | | | An | alysis | | | | | | Analys | s Set | | | Table Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | A1.1<br>A1.2<br>A1.3 | Part<br>A<br>1 | | A3.1 | A3.2 | | A5 | A6 | A7 | All<br>subjects | (B)<br>SAF | (B)<br>FAS | (B)<br>PPAS | Legend | Content | Overall and by age cohort |
| 1 | х | х | х | х | х | х | х | х | х | х | | | | Subject Overview | <ul> <li>Randomized subjects</li> <li>[Booster] Safety Analysis Set</li> <li>[Booster] Full Analysis Set</li> <li>[Booster] Per-Protocol Analysis Set</li> </ul> | х |
| 2 | Х | х | х | х | х | х | х | х | х | | х | Х | х | Subjects by Study Group<br>and Overall ([Population<br>Label]) | <ul> <li>Age cohort (only applicable for overall)</li> <li>B.b. s.l. serostatus at Screening</li> <li>B.b. s.l. serostatus at Month 18 (only applicable in Part B)</li> <li>Study Site</li> </ul> | х |
| 3 | Х | х | х | х | х | х | Х | х | х | | х | х | Х | Subjects by Visit ([Population Label]) | Incl. information whether visits were performed on site or remotely | Х |
| 4 | х | х | х | х | х | х | Х | х | Х | | х | Х | х | Attendance Status and<br>Early Termination<br>Details up to [Time<br>Point] ([Population<br>Label]) | <ul> <li>Number of early terminated subjects</li> <li>Primary reason for early termination</li> <li>All vaccinations administered</li> <li>Primary reason treatment discontinuation</li> <li>Individual stopping criteria</li> </ul> | х |

| | | | | Ana | alysis | | | | | | Analys | is Set | | | Table Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | A1.1<br>A1.2<br>A1.3 | Part<br>A<br>1 | | A3.1 | A3.2 | A4 | A5 | A6 | A7 | All<br>subjects | (B)<br>SAF | (B)<br>FAS | (B)<br>PPAS | Legend | Content | Overall<br>and by<br>age<br>cohort |
| 5 | x | x | x | x | x | x | x | x | x | | x | x | x | Vaccination Details<br>([Population Label]) | <ul> <li>Missed any vaccination</li> <li>Received only one vaccination</li> <li>Received only two vaccinations</li> <li>Received all three primary vaccinations (applicable for A1.1-A.3.1)</li> <li>1st vaccination performed</li> <li>2nd vaccination performed</li> <li>3rd vaccination performed</li> <li>Booster vaccination performed (applicable if A.3.2-A.7)</li> </ul> | X |
| 6 | х | Х | х | х | х | х | Х | х | х | | x | х | x | Protocol Deviations by<br>Deviation Type<br>([Population Label]) | <ul> <li>Subjects with relevant PDs</li> <li>Relevant PDs by category</li> <li>Subjects with not relevant PDs</li> <li>Not relevant PDs by category</li> <li>Major Monitor PDs</li> <li>Major Monitor PDs by category</li> <li>Minor Monitor PDs</li> <li>Minor Monitor PDs by category</li> </ul> | Х |
| 7 | Х | х | х | Х | х | х | Х | х | х | х | | | | Number of Screening<br>Failures and Reasons | <ul><li>Number of screening failures</li><li>Primary reason for screening failure</li></ul> | х |

#### 7.1.2 Baseline Evaluation

| | | | | Ana | lysis | | | | | An | alysis | Set | Tabl | e Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Parl | t A | | | Pa | art B | | | | | | | | Overall |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | (B)<br>SAF | (B)<br>FAS | (B)<br>PPAS | Legend | Content | and by<br>age<br>cohort |
| 1 | х | x | x | X | X | x | x | x | x | x | X | х | Summary Table of Demographic Data<br>([Population Label]) | <ul> <li>Gender</li> <li>Females with child-bearing potential</li> <li>Race</li> <li>Ethnicity</li> <li>Age at screening [years]</li> <li>Body height [cm]</li> <li>Body weight [kg]</li> <li>BMI [kg/m²]</li> </ul> | х |
| 2 | Х | х | х | х | х | х | х | х | х | х | х | Х | ECG Results at Screening ([Population Label]) | <ul><li>ECG result</li><li>Clinically relevant (if abnormal)</li></ul> | х |
| 3 | Х | х | х | х | х | х | х | х | х | х | х | Х | Medical History Overall and by SOC and PT ([Population Label]) | | х |
| 4 | Х | х | х | х | х | х | х | х | х | х | х | Х | Medical History Ongoing at Day 1<br>Overall and by SOC and PT<br>([Population Label]) | | х |
| 5 | Х | х | х | х | х | х | х | х | х | х | х | Х | Prior Medications Overall and by ATC<br>Level 2 and ATC Level 3 ([Population<br>Label]) | | х |
| 6 | Х | х | х | х | х | х | х | х | х | х | Х | Х | Concomitant Medications up to [Time Point] Overall and by ATC Level 2 and ATC Level 3 ([Population Label]) | | х |
| 7 | Х | х | Х | х | х | х | х | х | х | х | х | Х | Prior Procedures Overall and by SOC and PT ([Population Label]) | | х |
| 8 | Х | х | х | х | х | х | х | х | х | Х | Х | х | Concomitant Procedures up to [Time Point] Overall and by SOC and PT ([Population Label]) | | х |
| 9 | Х | х | х | Х | Х | Х | х | Х | Х | Х | Х | Х | Vaccination History Overall by ATC<br>Level 3 ([Population Label]) | | х |

Adapted from:
STAT03\_A Statistical Analysis Plan
Confidential and intellectual property of without prior written consent of


# 7.1.3 Immunogenicity Analysis

| | | | | Anal | ysis | | | | | Analy | sis Set | Table Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | | Part | Α | | | Pa | art B | 3 | | (D) | (D) | | Overall |
| טו | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4<br>3 | A5 | A6 | A7 | (B)<br>FAS | (B)<br>PPAS | Legend | and by<br>age<br>cohort |
| 1 | Х | х | х | х | х | х | х | х | х | | х | Number of Immunogenicity Blood Samples by Visit ([Population Label]) | |
| 2 | Х | х | х | х | х | х | х | х | Х | | х | ELISA: Number of Immunogenicity Results by OspA Specific Serotype ([Population Label]) | |
| 3 | Х | х | х | х | Х | Х | х | х | Х | х | х | ELISA: Number and Percentage of Subjects with OspA IgG Antibody Seropositive by Visit and OspA serotype ([Population Label]) | Х |
| 4 | Х | х | х | х | Х | Х | х | х | Х | х | х | ELISA: GMTs for OspA ST1 Specific IgG Antibodies by Visit ([Population Label]) | Х |
| 5 | Х | Х | х | х | Х | Х | х | х | Х | х | х | ELISA: GMTs for OspA ST2 Specific IgG Antibodies by Visit ([Population Label]) | Х |
| 6 | Х | х | х | х | Х | Х | х | Х | Х | х | х | ELISA: GMTs for OspA ST3 Specific IgG Antibodies by Visit ([Population Label]) | Х |
| 7 | Х | Х | х | х | Х | Х | х | Х | Х | х | х | ELISA: GMTs for OspA ST4 Specific IgG Antibodies by Visit ([Population Label]) | Х |
| 8 | Х | Х | х | х | Х | Х | х | Х | Х | х | х | ELISA: GMTs for OspA ST5 Specific IgG Antibodies by Visit ([Population Label]) | Х |
| 9 | Х | х | х | х | х | х | х | х | х | Х | Х | ELISA: GMTs for OspA ST6 Specific IgG Antibodies by Visit ([Population Label]) | Х |
| 10 | Х | х | х | х | х | х | х | х | х | | Х | ELISA: GMFRs (as compared to V0) for OspA ST1 Specific IgG<br>Antibodies by Visit ([Population Label]) | Х |
| 11 | Х | х | х | х | х | х | х | х | х | | х | ELISA: GMFRs (as compared to V0) for OspA ST2 Specific IgG<br>Antibodies by Visit ([Population Label]) | Х |
| 12 | Х | х | х | х | х | Х | х | х | Х | | х | ELISA: GMFRs (as compared to V0) for OspA ST3 Specific IgG<br>Antibodies by Visit ([Population Label]) | Х |
| 13 | х | х | Х | х | х | Х | Х | х | х | | х | ELISA: GMFRs (as compared to V0) for OspA ST4 Specific IgG Antibodies by Visit ([Population Label]) | Х |




| | | | | Anal | ysis | | | | | Analys | sis Set | Table Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | | Part | Α | | | P | art B | 3 | | (B) | (B) | | Overall and by |
| טו | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | <b>A4</b><br>3 | A5 | A6 | A7 | FAS | PPAS | Legend | age<br>cohort |
| 14 | Х | х | х | Х | х | х | х | х | х | | х | ELISA: GMFRs (as compared to V0) for OspA ST5 Specific IgG Antibodies by Visit ([Population Label]) | х |
| 15 | Х | х | х | х | х | х | х | х | х | | х | ELISA: GMFRs (as compared to V0) for OspA ST6 Specific IgG Antibodies by Visit ([Population Label]) | х |
| 16 | | | | | х | х | х | х | х | | х | ELISA: GMFRs (as compared to Day 208) for OspA ST1 Specific IgG Antibodies by Visit ([Population Label]) | х |
| 17 | | | | | Х | Х | Х | Х | Х | | х | ELISA: GMFRs (as compared to Day 208) for OspA ST2 Specific IgG Antibodies by Visit ([Population Label]) | х |
| 18 | | | | | Х | х | х | х | х | | х | ELISA: GMFRs (as compared to Day 208) for OspA ST3 Specific IgG Antibodies by Visit ([Population Label]) | Х |
| 19 | | | | | х | х | х | х | х | | х | ELISA: GMFRs (as compared to Day 208) for OspA ST4 Specific IgG Antibodies by Visit ([Population Label]) | х |
| 20 | | | | | х | х | Х | Х | х | | х | ELISA: GMFRs (as compared to Day 208) for OspA ST5 Specific IgG Antibodies by Visit ([Population Label]) | х |
| 21 | | | | | Х | Х | Х | Х | Х | | х | ELISA: GMFRs (as compared to Day 208) for OspA ST6 Specific IgG Antibodies by Visit ([Population Label]) | х |
| 22 | | | | | х | х | х | х | х | | х | ELISA: GMFRs (as compared to Day 365) for OspA ST1 Specific IgG Antibodies by Visit ([Population Label]) | х |
| 23 | | | | | х | х | х | х | х | | х | ELISA: GMFRs (as compared to Day 365) for OspA ST2 Specific IgG Antibodies by Visit ([Population Label]) | х |
| 24 | | | | | х | х | х | х | х | | х | ELISA: GMFRs (as compared to Day 365) for OspA ST3 Specific IgG Antibodies by Visit ([Population Label]) | х |
| 25 | | | | | х | х | х | х | х | | х | ELISA: GMFRs (as compared to Day 365) for OspA ST4 Specific IgG Antibodies by Visit ([Population Label]) | х |
| 26 | | | | | х | х | х | х | х | | х | ELISA: GMFRs (as compared to Day 365) for OspA ST5 Specific IgG Antibodies by Visit ([Population Label]) | х |
| 27 | | | | | х | х | х | х | х | | х | ELISA: GMFRs (as compared to Day 365) for OspA ST6 Specific IgG Antibodies by Visit ([Population Label]) | Х |
| 28 | | | | | Х | Х | х | х | х | | Х | ELISA: GMFRs (as compared to Month 18) for OspA ST1 Specific IgG Antibodies by Visit ([Population Label]) | Х |

| | | | | Anal | ysis | | | | | Analys | sis Set | Table Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | | Part | Α | | | P | art B | 3 | , | (B) | (B) | | Overall and by |
| | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4<br>3 | A5 | A6 | A7 | FAS | PPAS | Legend | age<br>cohort |
| 29 | | | | | х | х | х | х | х | | х | ELISA: GMFRs (as compared to Month 18) for OspA ST2 Specific IgG Antibodies by Visit ([Population Label]) | х |
| 30 | | | | | х | х | х | х | х | | х | ELISA: GMFRs (as compared to Month 18) for OspA ST3 Specific IgG Antibodies by Visit ([Population Label]) | х |
| 31 | | | | | х | | х | х | х | | х | ELISA: GMFRs (as compared to Month 18) for OspA ST4 Specific IgG Antibodies by Visit ([Population Label]) | х |
| 32 | | | | | х | х | х | х | х | | х | ELISA: GMFRs (as compared to Month 18) for OspA ST5 Specific IgG Antibodies by Visit ([Population Label]) | х |
| 33 | | | | | х | х | х | х | х | | х | ELISA: GMFRs (as compared to Month 18) for OspA ST6 Specific IgG Antibodies by Visit ([Population Label]) | х |
| 34 | Х | х | х | х | х | х | х | х | х | х | х | ELISA: Seroconversion Rate for OspA ST1 Specific IgG Antibodies by Visit ([Population Label]) | х |
| 35 | Х | х | х | х | х | х | х | х | х | х | х | ELISA: Seroconversion Rate for OspA ST2 Specific IgG Antibodies by Visit ([Population Label]) | х |
| 36 | Х | х | х | х | х | х | х | х | х | х | х | ELISA: Seroconversion for OspA ST3 Specific IgG Antibodies by Visit ([Population Label]) | х |
| 37 | Х | х | х | х | х | х | х | х | х | х | х | ELISA: Seroconversion Rate for OspA ST4 Specific IgG Antibodies by Visit ([Population Label]) | х |
| 38 | Х | х | х | х | х | х | х | х | х | х | х | ELISA: Seroconversion Rate for OspA ST5 Specific IgG Antibodies by Visit ([Population Label]) | х |
| 39 | Х | х | х | х | х | х | х | х | х | х | х | ELISA: Seroconversion Rate for OspA ST6 Specific IgG Antibodies by Visit ([Population Label]) | х |
| 40 | Х | х | х | х | х | х | х | х | х | | х | ELISA: Seroconversion Rate for OspA Specific IgG Antibodies against OspA Specific Serotypes ST1 to ST6 Combined by Visit ([Population Label]) | х |
| 41 | Х | х | х | х | х | х | х | х | х | | х | ELISA: Seroconversion Rate for OspA Specific IgG Antibodies against ST1 and ST2 Combined by Visit ([Population Label]) | Х |
| 42 | Х | х | х | х | х | Х | х | Х | х | Х | Х | ELISA: ANOVA (Factors: Study Group, Age Cohort <sup>4</sup> ) for GMT of OspA ST1 Specific IgG Antibodies by Visit ([Population Label]) | |

<sup>&</sup>lt;sup>4</sup> For Interim Analysis 1.1, age group will be not used as factor for ANOVA.

Adapted from:

STATO3\_A Statistical Analysis Plan Version 6.0, Effective Date 16-Feb-2018

without prior written consent of

| | | | | Anal | ysis | | | | | Analys | sis Set | Table Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | | Part | Α | | | Pa | art B | 3 | | (B) | (B) | | Overall and by |
| | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4<br>3 | A5 | A6 | A7 | FAS | PPAS | Legend | age<br>cohort |
| 43 | Х | х | х | х | х | х | х | х | х | х | х | ELISA: ANOVA (Factors: Study Group, Age Cohort <sup>4</sup> ) for GMT of OspA ST2 Specific IgG Antibodies by Visit ([Population Label]) | |
| 44 | Х | Х | х | х | Х | Х | х | х | х | х | х | ELISA: ANOVA (Factors: Study Group, Age Cohort <sup>4</sup> ) for GMT of OspA ST3 Specific IgG Antibodies by Visit ([Population Label]) | |
| 45 | Х | х | х | х | х | х | х | х | х | х | Х | ELISA: ANOVA (Factors: Study Group, Age Cohort <sup>4</sup> ) for GMT of OspA ST4 Specific IgG Antibodies by Visit ([Population Label]) | |
| 46 | Х | х | х | х | х | х | х | х | х | х | Х | ELISA: ANOVA (Factors: Study Group, Age Cohort <sup>4</sup> ) for GMT of OspA ST5 Specific IgG Antibodies by Visit ([Population Label]) | |
| 47 | Х | Х | х | х | Х | х | х | х | х | х | Х | ELISA: ANOVA (Factors: Study Group, Age Cohort <sup>4</sup> ) for GMT of OspA ST6 Specific IgG Antibodies by Visit ([Population Label]) | |
| 48 | Х | х | х | х | х | Х | х | х | х | х | х | ELISA: ANOVA (Factors: Study Group, Study Site, Age Cohort, Age Cohort*Study Group and Baseline B.b. s.l. Serostatus <sup>4</sup> ) for GMT of OspA ST1 Specific IgG Antibodies by Visit ([Population Label]) | |
| 49 | Х | х | х | х | х | х | х | х | х | х | х | ELISA: ANOVA (Factors: Study Group, Study Site, Age Cohort, Age Cohort*Study Group and Baseline B.b. s.l. Serostatus <sup>4</sup> ) for GMT of OspA ST2 Specific IgG Antibodies by Visit ([Population Label]) | |
| 50 | х | х | х | х | х | х | х | х | х | х | х | ELISA: ANOVA (Factors: Study Group, Study Site, Age Cohort, Age Cohort*Study Group, and Baseline B.b. s.l. Serostatus <sup>4</sup> ) for GMT of OspA ST3 Specific IgG Antibodies by Visit ([Population Label]) | |
| 51 | х | х | х | х | х | х | х | х | х | х | х | ELISA: ANOVA (Factors: Study Group, Study Site, Age Cohort, Age Cohort*Study Group and Baseline B.b. s.l. Serostatus <sup>4</sup> ) for GMT of OspA ST4 Specific IgG Antibodies by Visit ([Population Label]) | |
| 52 | х | х | х | х | х | х | х | х | х | х | х | ELISA: ANOVA (Factors: Study Group, Study Site, Age Cohort, Age Cohort*Study Group and Baseline B.b. s.l. Serostatus <sup>4</sup> ) for GMT of OspA ST5 Specific IgG Antibodies by Visit ([Population Label]) | |
| 53 | Х | х | х | х | х | Х | х | х | х | х | х | ELISA: ANOVA (Factors: Study Group, Study Site, Age Cohort, Age Cohort*Study Group and Baseline B.b. s.l. Serostatus <sup>4</sup> ) for GMT of OspA ST6 Specific IgG Antibodies by Visit ([Population Label]) | |
| 54 | х | х | х | х | | | | | | | х | ELISA: ANOVA (Factors: Study Group, Age Cohort <sup>4</sup> ) for GMFR from Screening at Day 208 of OspA ST1 Specific IgG Antibodies ([Population Label]) | |

| | | | | Anal | lysis | | | | | Analy | sis Set | Table Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | | Part | Α | Part B 2 A3.1 A3.2 A4 A5 A6 A | | | (B) | (B) | | Overall and by | | | |
| l l | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | <b>A4</b> 3 | A5 | A6 | A7 | FAS | PPAS | Legend | age<br>cohort |
| | | | | | х | х | х | х | х | | х | ELISA: ANOVA (Factors: Study Group, Age Cohort <sup>4</sup> ) for GMFR from<br>Screening at Day 208 and Month 19 of OspA ST1 Specific IgG<br>Antibodies ([Population Label]) | |
| 55 | Х | х | х | х | | | | | | | х | ELISA: ANOVA (Factors: Study Group, Age Cohort <sup>4</sup> ) for GMFR from Screening at Day 208 of OspA ST2 Specific IgG Antibodies ([Population Label]) | |
| | | | | | х | х | х | х | х | | х | ELISA: ANOVA (Factors: Study Group, Age Cohort <sup>4</sup> ) for GMFR from<br>Screening at Day 208 and Month 19 of OspA ST2 Specific IgG<br>Antibodies ([Population Label]) | |
| 56 | Х | х | х | х | | | | | | | х | ELISA: ANOVA (Factors: Study Group, Age Cohort <sup>4</sup> ) for GMFR from<br>Screening at Day 208 of OspA ST3 Specific IgG Antibodies<br>([Population Label]) | |
| | | | | | х | х | х | х | х | | х | ELISA: ANOVA (Factors: Study Group, Age Cohort <sup>4</sup> ) for GMFR from<br>Screening at Day 208 and Month 19 of OspA ST3 Specific IgG<br>Antibodies ([Population Label]) | |
| 57 | Х | х | х | х | | | | | | | х | ELISA: ANOVA (Factors: Study Group, Age Cohort <sup>4</sup> ) for GMFR from<br>Screening at Day 208 of OspA ST4 Specific IgG Antibodies<br>([Population Label]) | |
| 31 | | | | | х | х | х | х | х | | х | ELISA: ANOVA (Factors: Study Group, Age Cohort <sup>4</sup> ) for GMFR from<br>Screening at Day 208 and Month 19 of OspA ST4 Specific IgG<br>Antibodies ([Population Label]) | |
| 58 | Х | х | х | х | | | | | | | х | ELISA: ANOVA (Factors: Study Group, Age Cohort <sup>4</sup> ) for GMFR from Screening at Day 208 of OspA ST5 Specific IgG Antibodies ([Population Label]) | |
| 55 | | | | | х | х | х | х | х | | х | ELISA: ANOVA (Factors: Study Group, Age Cohort <sup>4</sup> ) for GMFR from<br>Screening at Day 208 and Month 19 of OspA ST5 Specific IgG<br>Antibodies ([Population Label]) | |
| 59 | Х | х | х | х | | | | | | | Х | ELISA: ANOVA (Factors: Study Group, Age Cohort <sup>4</sup> ) for GMFR from<br>Screening at Day 208 of OspA ST6 Specific IgG Antibodies<br>([Population Label]) | |

| | | | | Anal | ysis | | | | | Analys | sis Set | Table Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | | Part | Α | 1 | | P | art B | } | , | (B) | (B) | | Overall and by |
| | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4<br>3 | A5 | A6 | A7 | FAS | PPAS | Legend | age<br>cohort |
| | | | | | х | х | х | х | х | | x | ELISA: ANOVA (Factors: Study Group, Age Cohort <sup>4</sup> ) for GMFR from<br>Screening at Day 208 and Month 19 of OspA ST6 Specific IgG<br>Antibodies ([Population Label]) | |
| 60 | Х | х | х | х | | | | | | x | х | ELISA: ANOVA (Factors: Study Group, Study Site, Age Cohort, Age Cohort*Study Group and Baseline B.b. s.l. Serostatus <sup>4</sup> ) for GMFR from Screening at Day 208 of OspA ST1 Specific IgG Antibodies ([Population Label]) | |
| 00 | | | | | х | х | х | х | Х | | x | ELISA: ANOVA (Factors: Study Group, Study Site, Age Cohort, Age Cohort*Study Group and Baseline B.b. s.l. Serostatus <sup>4</sup> ) for GMFR from Screening at Day 208 and Month 19 of OspA ST1 Specific IgG Antibodies ([Population Label]) | |
| 61 | Х | х | х | х | | | | | | | х | ELISA: ANOVA (Factors: Study Group, Study Site, Age Cohort, Age Cohort*Study Group and Baseline B.b. s.l. Serostatus <sup>4</sup> ) for GMFR from Screening at Day 208 of OspA ST2 Specific IgG Antibodies ([Population Label]) | |
| 01 | | | | | х | х | х | х | Х | | х | ELISA: ANOVA (Factors: Study Group, Study Site, Age Cohort, Age Cohort*Study Group and Baseline B.b. s.l. Serostatus <sup>4</sup> ) for GMFR from Screening at Day 208 and Month 19 of OspA ST2 Specific IgG Antibodies ([Population Label]) | |
| 62 | Х | х | х | х | | | | | | | х | ELISA: ANOVA (Factors: Study Group, Study Site, Age Cohort, Age Cohort*Study Group and Baseline B.b. s.l. Serostatus <sup>4</sup> ) for GMFR from Screening at Day 208 of OspA ST3 Specific IgG Antibodies ([Population Label]) | |
| 02 | | | | | х | х | х | х | Х | | х | ELISA: ANOVA (Factors: Study Group, Study Site, Age Cohort, Age Cohort*Study Group and Baseline B.b. s.l. Serostatus <sup>4</sup> ) for GMFR from Screening at Day 208 and Month 19 of OspA ST3 Specific IgG Antibodies ([Population Label]) | |
| 63 | Х | х | х | Х | | | | | | | х | ELISA: ANOVA (Factors: Study Group, Study Site, Age Cohort, Age Cohort*Study Group and Baseline B.b. s.l. Serostatus <sup>4</sup> ) for GMFR from Screening at Day 208 of OspA ST4 Specific IgG Antibodies ([Population Label]) | |

| | | | | Anal | ysis | | | | | Analys | sis Set | Table Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | | Part | Α | 1 | Part B A3.2 A4 A5 A6 A7 | | | (B) | (B) | | Overall and by | | |
| | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4<br>3 | A5 | A6 | A7 | FAS | PPAS | Legend | age<br>cohort |
| | | | | | х | х | х | х | Х | | х | ELISA: ANOVA (Factors: Study Group, Study Site, Age Cohort, Age Cohort*Study Group and Baseline B.b. s.l. Serostatus <sup>4</sup> ) for GMFR from Screening at Day 208 and Month 19 of OspA ST4 Specific IgG Antibodies ([Population Label]) | |
| 64 | Х | х | х | Х | | | | | | X | ELISA: ANOVA (Factors: Study Group, Study Site, Age Cohort, Age Cohort*Study Group and Baseline B.b. s.l. Serostatus <sup>4</sup> ) for GMFR from Screening at Day 208 of OspA ST5 Specific IgG Antibodies ([Population Label]) | | |
| 04 | | | | | х | х | х | Х | X | | x | ELISA: ANOVA (Factors: Study Group, Study Site, Age Cohort, Age Cohort*Study Group and Baseline B.b. s.l. Serostatus <sup>4</sup> ) for GMFR from Screening at Day 208 and Month 19 of OspA ST5 Specific IgG Antibodies ([Population Label]) | |
| 65 | Х | х | х | х | | | | | | | x | ELISA: ANOVA (Factors: Study Group, Study Site, Age Cohort, Age Cohort*Study Group and Baseline B.b. s.l. Serostatus <sup>4</sup> ) for GMFR from Screening at Day 208 of OspA ST6 Specific IgG Antibodies ([Population Label]) | |
| 03 | | | | | х | х | х | х | Х | | х | ELISA: ANOVA (Factors: Study Group, Study Site, Age Cohort, Age Cohort*Study Group and Baseline B.b. s.l. Serostatus <sup>4</sup> ) for GMFR from Screening at Day 208 and Month 19 of OspA ST6 Specific IgG Antibodies ([Population Label]) | |
| | Х | х | х | х | | | | | | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST1 vs ST2 at Day 208 ([Population Label]) | |
| 66 | | | | | х | х | х | х | Х | | Х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST1 vs ST2 at Day 208 and Month 19 ([Population<br>Label]) | |
| | Х | х | х | х | | | | | | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST1 vs ST3 at Day 208 ([Population Label]) | |
| 67 | | | | | х | х | х | х | х | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST1 vs ST3 at Day 208 and Month 19 ([Population<br>Label]) | |
| 68 | Х | х | х | х | | | | | | | Х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST1 vs ST4 at Day 208 ([Population Label]) | S of 110 |

Adapted from: STAT03\_A Statistical Analysis Plan Version 6.0, Effective Date 16-Feb-2018

without prior written consent of


| | | | | Anal | ysis | | | | | Analys | sis Set | Table Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | | Part | Α | 1 | | P | art B | 3 | , | (B) | (B) | | Overall and by |
| | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4<br>3 | A5 | A6 | A7 | FAS | PPAS | Legend | age<br>cohort |
| | | | | | х | х | х | х | х | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST1 vs ST4 at Day 208 and Month 19 ([Population<br>Label]) | |
| | Х | Х | х | х | | | | | | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST1 vs ST5 at Day 208 ([Population Label]) | |
| 69 | | | | | х | х | х | х | х | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST1 vs ST5 Day 208 and Month 19 ([Population<br>Label]) | |
| | Х | х | х | х | | | | | | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST1 vs ST6 at Day 208 ([Population Label]) | |
| 70 | | | | | х | х | х | х | х | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST1 vs ST6 at Day 208 and Month 19 ([Population<br>Label]) | |
| | Х | х | х | х | | | | | | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST2 vs ST3 at Day 208 ([Population Label]) | |
| 71 | | | | | х | х | х | х | х | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST2 vs ST3 at Day 208 and Month 19 ([Population<br>Label]) | |
| | Х | х | х | х | | | | | | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST2 vs ST4 at Day 208 ([Population Label]) | |
| 72 | | | | | х | х | х | х | х | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST2 vs ST4 at Day 208 and Month 19 ([Population<br>Label]) | |
| | Х | х | х | х | | | | | | | Х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST2 vs ST5 at Day 208 ([Population Label]) | |
| 73 | | | | | х | х | х | х | х | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST2 vs ST5 at Day 208 and Month 19 ([Population<br>Label]) | |
| 74 | х | х | Х | Х | | | | | | | Х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST2 vs ST6 at Day 208 ([Population Label]) | |

| | | | | Anal | ysis | | | | | Analys | sis Set | Table Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | | Part | Α | 1 | | P | art B | } | , | (B) | (B) | | Overall and by |
| | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4<br>3 | A5 | A6 | A7 | FAS | PPAS | Legend | age<br>cohort |
| | | | | | х | х | х | х | х | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST2 vs ST6 at Day 208 and Month 19 ([Population<br>Label]) | |
| | Х | Х | х | Х | | | | | | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST3 vs ST4 at Day 208 ([Population Label]) | |
| 75 | | | | | х | х | х | х | х | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST3 vs ST4 at Day 208 and Month 19 ([Population<br>Label]) | |
| | Х | Х | х | | | | | | | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST3 vs ST5 at Day 208 ([Population Label]) | |
| 76 | | | | | х | Х | х | х | х | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST3 vs ST5 at Day 208 and Month 19 ([Population<br>Label]) | |
| | Х | х | х | х | | | | | | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST3 vs ST6 at Day 208 ([Population Label]) | |
| 77 | | | | | х | Х | х | х | х | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST3 vs ST6 at Day 208 and Month 19 ([Population<br>Label]) | |
| | Х | Х | х | х | | | | | | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST4 vs ST5 at Day 208 ([Population Label]) | |
| 78 | | | | | х | Х | х | х | х | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST4 vs ST5 at Day 208 and Month 19 ([Population<br>Label]) | |
| | Х | х | х | х | | | | | | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST4 vs ST6 at Day 208 ([Population Label]) | |
| 79 | | | | | х | х | х | х | х | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST4 vs ST6 at Day 208 and Month 19 ([Population<br>Label]) | |
| 80 | х | х | х | х | | | | | | | Х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST5 vs ST6 at Day 208 ([Population Label]) | |

| | | | | Anal | ysis | | | | | Analys | sis Set | Table Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | | Part | Α | 1 | | P | art B | } | , | (B) | (B) | | Overall and by |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4<br>3 | A5 | A6 | A7 | FAS | PPAS | Legend | age<br>cohort |
| | | | | | х | х | х | х | х | | х | ELISA: Correlation Analysis for GMTs of OspA Specific IgG<br>Antibodies for ST5 vs ST6 at Day 208 and Month 19 ([Population<br>Label]) | |
| CCI | | | 1 | | | 1 | 1 | | | | | | |




Adapted from:
STAT03\_A Statistical Analysis Plan

without prior written consent of




Adapted from:
STAT03\_A Statistical Analysis Plan

without prior written consent of













Adapted from:

STATO3\_A Statistical Analysis Plan Version 6.0, Effective Date 16-Feb-2018

without prior written consent of

Confidential and intellectual property of \_\_\_\_\_. No part of this document or its contents may be duplicated, referenced, published or otherwise disclosed in any form or by any means





| | | | | Anal | ysis | | | | | Analys | is Set | Table Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 15 | I | Part | Α | | | P | art B | } | | (D) | (D) | | Overall |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4<br>3 | A5 | A6 | A7 | (B)<br>FAS | (B)<br>PPAS | Legend | and by<br>age<br>cohort |
| | | | | | | | | | | | | CCI | |
| 159 | | | | | | | | | | | | | |
| | | | | | - | - | | | | | _ | | |
| 1 | | l | | | | | | | | | | | 1 |

# 7.1.4 Adverse Events

| | | | | | Aı | nalysis | | | | | 1 | Table Description | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sub | | Part | Α | 1 | | 1 | Part B | 1 | 1 | | | Overall | Including |
| ID | -ID | A1.1<br>A1.2 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content | and by age | statistical<br>test |
| Solic | ited a | A1.3<br>nd Unsoli | cited A | dverse | Fvent | 9 | | | | | | | cohort | |
| 1 | ited al | X | x | X | X | x | x | x | x | x | Summary Table of Adverse Events<br>up to [Time Point] (solicited and<br>unsolicited) ([Booster] Safety<br>Analysis Set) | Any AE, related AE, severe AE, related severe AE, related SAE, medically attended AE, related medically attended AE, AE leading to withdrawal from study, AE leading to withdrawal from further vaccination Any solicited AE, severe solicited AE, solicited local AE, solicited local AE, solicited | x | x |

| | | | | | Ar | nalysis | | | | | 1 | able Description | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sub | | Part | Α | , | | | Part B | | | | | Overall | Including |
| ID | -ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content | and by<br>age<br>cohort | statistical<br>test |
| | | | | | | | | | | | | systemic AE, severe solicited systemic AE • Any unsolicited AE, related unsolicited AE, severe unsolicited AE, related severe unsolicited AE, unsolicited SAE, medically attended unsolicited AE, related medically attended unsolicited AE, unsolicited AE leading to withdrawal from study, unsolicited AE leading to withdrawal from further vaccination, AEs of special interest, related AEs of special interest | | |
| 2 | 1 | Х | Х | х | х | х | Х | Х | Х | Х | Summary Table of Adverse Events<br>up to [Time Point] by Vaccination<br>Period (solicited and unsolicited)<br>([Booster] Safety Analysis Set) | see Table ID 1 | Х | х |
| 2 | 2 | Х | х | х | х | х | х | х | х | х | Summary Table of Adverse Events<br>up to [Time Point] after first<br>Vaccination (solicited and<br>unsolicited) ([Booster] Safety<br>Analysis Set) | see Table ID 1 | Х | Х |
| 2 | 3 | х | х | х | х | х | х | х | х | х | Summary Table of Adverse Events<br>up to [Time Point] after second<br>Vaccination (solicited and<br>unsolicited) ([Booster] Safety<br>Analysis Set) | see Table ID 1 | х | х |


| | | | | | Ar | nalysis | | | | | T | able Description | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sub | | Part | Α | | | | Part B | | | | | Overall | Including |
| ID | -ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content | and by<br>age<br>cohort | statistical<br>test |
| 2 | 4 | X | х | x | x | x | х | х | х | х | Summary Table of Adverse Events<br>up to [Time Point] after third<br>Vaccination (solicited and<br>unsolicited) ([Booster] Safety<br>Analysis Set) | see Table ID 1 | х | х |
| 2 | 5 | | | | | х | х | х | х | х | Summary Table of Adverse Events<br>up to [Time Point] after Booster<br>Vaccination (solicited and<br>unsolicited) (Booster Safety<br>Analysis Set) | see Table ID 1 | х | х |
| 3 | | Х | Х | Х | х | х | х | х | х | х | Solicited and Unsolicited Serious<br>Adverse Events up to [Time Point]<br>by SOC and PT ([Booster] Safety<br>Analysis Set) | | х | х |
| 4 | | х | х | х | х | х | х | х | х | х | Solicited and Unsolicited Related<br>Serious Adverse Events up to<br>[Time Point] by SOC and PT<br>([Booster] Safety Analysis Set) | | х | х |
| 5 | | х | х | х | х | х | х | х | х | х | Solicited and Unsolicited Medically<br>Attended Adverse Events up to<br>[Time Point] by SOC and PT<br>([Booster] Safety Analysis Set) | | х | х |
| 6 | | Х | х | х | х | х | х | х | х | х | Solicited and Unsolicited Related<br>Medically Attended Adverse Events<br>up to [Time Point] by SOC and PT<br>([Booster] Safety Analysis Set) | | х | х |
| 7 | | X | х | | | | | | | | Solicited and Unsolicited Adverse<br>Events up to [Time Point] Leading<br>to Withdrawal from further<br>Vaccination by SOC and PT<br>([Booster] Safety Analysis Set) | | х | х |

| | | | | | Ar | nalysis | | | | | Т | able Description | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sub | | Part | Α | | | | Part B | | | | · | Overall | Including |
| ID | -ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content | and by<br>age<br>cohort | statistical<br>test |
| 8 | | Х | х | x | х | х | х | x | х | x | Solicited and Unsolicited Adverse<br>Events up to [Time Point] Leading<br>to Withdrawal from Study by SOC<br>and PT ([Booster] Safety Analysis<br>Set) | | х | Х |
| 9 | | х | Х | х | х | х | Х | Х | х | х | Any Non-Serious Adverse Events<br>up to [Time Point] by SOC and PT<br>for PTs with Frequency >5% in any<br>Study Group (eCRF Section 'AE<br>Log' for Unsolicited AEs and<br>'Subject Diary' for Solicited AEs,<br>[Booster] Safety Analysis Set) | <ul><li>Overall</li><li>Solicited</li><li>Unsolicited</li></ul> | x | х |
| 10 | | х | Х | х | х | х | Х | Х | х | х | Any Non-Serious Adverse Events<br>up to [Time Point] by SOC and PT<br>for PTs with Frequency >10% in<br>any Study Group (eCRF Section 'AE<br>Log' for Unsolicited AEs and<br>'Subject Diary' for Solicited AEs,<br>([Booster] Safety Analysis Set) | <ul><li>Overall</li><li>Solicited</li><li>Unsolicited</li></ul> | Х | х |
| Solic | ited Ad | dverse Ev | /ents | | | | | | | , | | | | |
| 11 | | Х | х | | | х | | | | | Solicited Adverse Events after any<br>Vaccination ([Booster] Safety<br>Analysis Set) | <ul> <li>Any solicited AE</li> <li>Any solicited local AE</li> <li>Any solicited<br/>systemic AE</li> </ul> | х | Х |
| 12 | | Х | х | | | х | | | | | Severe Solicited Adverse Events<br>after any Vaccination by Symptom<br>([Booster] Safety Analysis Set) | | Х | Х |
| 13 | | х | х | | | х | | | | | Solicited Local Adverse Events<br>after any Vaccination by Symptom<br>([Booster] Safety Analysis Set) | <ul> <li>Any solicited local AE</li> <li>Any solicited local AE meeting FDA Grading Scale</li> </ul> | х | х |

Adapted from:
STAT03\_A Statistical Analysis Plan

without prior written consent of


| | | | | | A | nalysis | | | | | ] | able Description | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sub | | Part | Α | | | | Part B | | | | | Overall | Including |
| ID | -ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content | and by<br>age<br>cohort | statistical<br>test |
| | | | | | | | | | | | | Pain Tenderness Induration/hardening Induration/hardening Meeting FDA Grading Scale Swelling Swelling meeting FDA Grading Scale Erythema/ redness Erythema/ redness Frythema/ redness Meeting FDA Grading Scale Add footnote that different grading scales are applicable for the different age cohorts. | | |
| 14 | | x | х | | | х | | | | | Solicited Systemic Adverse Events after any Vaccination by Symptom ([Booster] Safety Analysis Set) Solicited Adverse Events after any | <ul> <li>Headache</li> <li>Muscle pain</li> <li>Joint pain</li> <li>Nausea</li> <li>Vomiting</li> <li>Fatigue</li> <li>Fever</li> </ul> | х | х |
| 15 | | Х | х | | | х | | | | | Vaccination - Classified by<br>Maximum Severity ([Booster]<br>Safety Analysis Set) | | Х | Х |
| 16 | | Х | Х | | | х | | | | | Solicited Local Adverse Events after any Vaccination by Symptom | | Х | Х |

| ID | | | | | Aı | nalysis | | | | | Ta | able Description | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sub<br>-ID | | Part B | | | | | | | Overall | los also altes et | | | |
| | | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content | and by<br>age<br>cohort | Including<br>statistical<br>test |
| | | | | | | | | | | | Classified by Maximum Severity<br>([Booster] Safety Analysis Set) | | | |
| 17 | | х | х | | | х | | | | | Solicited Systemic Adverse Events<br>after any Vaccination by Symptom<br>Classified by Maximum Severity<br>([Booster] Safety Analysis Set) | | х | х |
| 18 | 1 | х | х | | | х | | | | | Solicited Adverse Events by<br>Vaccination Period ([Booster]<br>Safety Analysis Set) | | х | х |
| 18 | 2 | х | х | | | х | | | | | Solicited Adverse Events after first<br>Vaccination ([Booster] Safety<br>Analysis Set) | | х | х |
| 18 | 3 | х | х | | | х | | | | | Solicited Adverse Events after<br>second Vaccination ([Booster]<br>Safety Analysis Set) | | х | х |
| 18 | 4 | х | х | | | х | | | | | Solicited Adverse Events after third<br>Vaccination ([Booster] Safety<br>Analysis Set) | | х | х |
| 18 | 5 | | | | | х | | | | | Solicited Adverse Events after<br>Booster Vaccination (Booster<br>Safety Analysis Set) | | х | х |
| 19 | 1 | х | х | | | х | | | | | Severe Solicited Adverse Events by<br>Symptom and Vaccination Period<br>([Booster] Safety Analysis Set) | | х | х |
| 19 | 2 | х | х | | | х | | | | | Severe Solicited Adverse Events by<br>Symptom after first vaccination<br>([Booster] Safety Analysis Set) | | х | х |
| 19 | 3 | х | х | | | х | | | | | Severe Solicited Adverse Events<br>after second Vaccination by<br>Symptom ([Booster] Safety<br>Analysis Set) | | х | х |

| ID | | | | | Aı | nalysis | | | | | Т | able Description | | nd by statistical age | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|--|--|
| | Sub<br>-ID | | Part B | | | | | | Overall | Including | | | | | | |
| | | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content | and by<br>age<br>cohort | statistical | | |
| 19 | 4 | х | х | | | х | | | | | Severe Solicited Adverse Events<br>after third Vaccination by Symptom<br>([Booster] Safety Analysis Set) | | х | х | | |
| 19 | 5 | | | | | х | | | | | Severe Solicited Adverse Events<br>after Booster Vaccination by<br>Symptom (Booster Safety Analysis<br>Set) | | х | х | | |
| 20 | 1 | х | х | | | х | | | | | Solicited Local Adverse Events by<br>Symptom and Vaccination Period<br>([Booster] Safety Analysis Set) | See Table ID 13 | х | х | | |
| 20 | 2 | х | х | | | х | | | | | Solicited Local Adverse Events<br>after first Vaccination by Symptom<br>([Booster] Safety Analysis Set) | See Table ID 13 | х | х | | |
| 20 | 3 | х | х | | | х | | | | | Solicited Local Adverse Events<br>after second Vaccination by<br>Symptom ([Booster] Safety<br>Analysis Set) | See Table ID 13 | х | х | | |
| 20 | 4 | х | х | | | х | | | | | Solicited Local Adverse Events<br>after third Vaccination by Symptom<br>([Booster] Safety Analysis Set) | See Table ID 13 | х | х | | |
| 20 | 5 | | | | | х | | | | | Solicited Local Adverse Events<br>after Booster Vaccination by<br>Symptom (Booster Safety Analysis<br>Set) | See Table ID 13 | х | х | | |
| 21 | 1 | х | х | | | х | | | | | Solicited Systemic Adverse Events<br>by Symptom and Vaccination<br>Period ([Booster] Safety Analysis<br>Set) | | х | х | | |
| 21 | 2 | Х | х | | | х | | | | | Solicited Systemic Adverse Events<br>after first Vaccination by Symptom<br>([Booster] Safety Analysis Set) | | Х | Х | | |
| | | | | | Ar | nalysis | | | | | Ta | able Description | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sub | | Part | Α | | | | Part B | | | | - | Overall | Including |
| ID | -ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content | and by<br>age<br>cohort | statistical<br>test |
| 21 | 3 | Х | х | | | х | | | | | Solicited Systemic Adverse Events<br>after second Vaccination by<br>Symptom ([Booster] Safety<br>Analysis Set) | | х | х |
| 21 | 4 | х | х | | | х | | | | | Solicited Systemic Adverse Events<br>after third Vaccination by Symptom<br>([Booster] Safety Analysis Set) | | х | x |
| 21 | 5 | | | | | х | | | | | Solicited Systemic Adverse Events<br>after Booster Vaccination by<br>Symptom (Booster Safety Analysis<br>Set) | | х | х |
| 22 | 1 | х | х | | | х | | | | | Solicited Adverse Events by Vaccination Period and Classified by Maximum Severity ([Booster] Safety Analysis Set) | | х | х |
| 22 | 2 | х | х | | | х | | | | | Solicited Adverse Events after first<br>Vaccination - Classified by<br>Maximum Severity ([Booster]<br>Safety Analysis Set) | | х | х |
| 22 | 3 | х | х | | | х | | | | | Solicited Adverse Events after<br>second Vaccination - Classified by<br>Maximum Severity ([Booster]<br>Safety Analysis Set) | | х | х |
| 22 | 4 | Х | Х | | | х | | | | | Solicited Adverse Events after third<br>Vaccination by Classified -<br>Maximum Severity ([Booster]<br>Safety Analysis Set) | | х | х |
| 22 | 5 | | | | | х | | | | | Solicited Adverse Events after Booster Vaccination - Classified by Maximum Severity (Booster Safety Analysis Set) | | х | х |


| | | | | | Ar | nalysis | | | | | Т | able Description | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sub | | Part | Α. | | | | Part B | | | | | Overall | Including |
| ID | -ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content | and by<br>age<br>cohort | statistical<br>test |
| 23 | 1 | Х | х | | | х | | | | | Solicited Local Adverse Events by<br>Symptom and Vaccination Period<br>Classified by Maximum Severity<br>([Booster] Safety Analysis Set) | | х | х |
| 23 | 2 | Х | х | | | х | | | | | Solicited Local Adverse Events<br>after first Vaccination by Symptom<br>Classified by Maximum Severity<br>([Booster] Safety Analysis Set) | | х | х |
| 23 | 3 | х | х | | | х | | | | | Solicited Local Adverse Events<br>after second Vaccination by<br>Symptom Classified by Maximum<br>Severity ([Booster] Safety Analysis<br>Set) | | х | х |
| 23 | 4 | х | х | | | х | | | | | Solicited Local Adverse Events<br>after third Vaccination by Symptom<br>Classified by Maximum Severity<br>([Booster] Safety Analysis Set) | | х | х |
| 23 | 5 | | | | | х | | | | | Solicited Local Adverse Events<br>after Booster Vaccination by<br>Symptom Classified by Maximum<br>Severity (Booster Safety Analysis<br>Set) | | Х | х |
| 24 | 1 | Х | х | | | х | | | | | Solicited Systemic Adverse Events<br>by Symptom and Vaccination<br>Period - Classified by Maximum<br>Severity ([Booster] Safety Analysis<br>Set) | | Х | х |
| 24 | 2 | х | х | | | х | | | | | Solicited Systemic Adverse Events<br>after first Vaccination by Symptom<br>Classified by Maximum Severity<br>([Booster] Safety Analysis Set) | | х | х |

| | | | | | Aı | nalysis | | | | | Ţ. | able Description | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sub | | Part | Α | | | | Part B | | | | | Overall | Including |
| ID | -ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content | and by<br>age<br>cohort | statistical<br>test |
| 24 | 3 | Х | х | | | х | | | | | Solicited Systemic Adverse Events<br>after second Vaccination by<br>Symptom Classified by Maximum<br>Severity ([Booster] Safety Analysis<br>Set) | | х | х |
| 24 | 4 | х | х | | | х | | | | | Solicited Systemic Adverse Events<br>after third Vaccination by Symptom<br>Classified by Maximum Severity<br>([Booster] Safety Analysis Set) | | х | х |
| 24 | 5 | | | | | х | | | | | Solicited Systemic Adverse Events<br>after Booster Vaccination by<br>Symptom Classified by Maximum<br>Severity (Booster Safety Analysis<br>Set) | | х | х |
| 25 | 1 | х | х | | | х | | | | | Solicited Adverse Events by Diary<br>Day and Vaccination Period<br>([Booster] Safety Analysis Set) | | х | х |
| 25 | 2 | х | х | | | х | | | | | Solicited Adverse Events after first<br>Vaccination by Diary Day ([Booster]<br>Safety Analysis Set) | | х | х |
| 25 | 3 | х | х | | | х | | | | | Solicited Adverse Events after<br>second Vaccination by Diary Day<br>([Booster] Safety Analysis Set) | | х | х |
| 25 | 4 | х | х | | | х | | | | | Solicited Adverse Events after third<br>Vaccination by Diary ([Booster]<br>Safety Analysis Set) | | х | х |
| 25 | 5 | | | | | х | | | | | Solicited Adverse Events after<br>Booster Vaccination by Diary Day<br>(Booster Safety Analysis Set) | | х | х |
| 26 | 1 | Х | х | | | х | | | | | Solicited Local Adverse Events by<br>Diary Day and Vaccination Period<br>([Booster] Safety Analysis Set) | | Х | х |


| | | | | | Aı | nalysis | | | | | T. | able Description | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sub | | Part | : A | | | | Part B | } | | | | Overall | Including |
| ID | -ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content | and by<br>age<br>cohort | statistical<br>test |
| 26 | 2 | х | х | | | х | | | | | Solicited Local Adverse Events<br>after first Vaccination by Diary Day<br>([Booster] Safety Analysis Set) | | х | х |
| 26 | 3 | х | х | | | х | | | | | Solicited Local Adverse Events<br>after second Vaccination by Diary<br>Day ([Booster] Safety Analysis Set) | | х | х |
| 26 | 4 | х | х | | | х | | | | | Solicited Local Adverse Events<br>after third Vaccination by Diary Day<br>([Booster] Safety Analysis Set) | | х | х |
| 26 | 5 | | | | | х | | | | | Solicited Local Adverse Events<br>after Booster Vaccination by Diary<br>Day (Booster Safety Analysis Set) | | х | х |
| 27 | 1 | х | х | | | х | | | | | Solicited Systemic Adverse Events<br>by Diary Day and Vaccination<br>Period ([Booster] Safety Analysis<br>Set) | | х | х |
| 27 | 2 | Х | х | | | х | | | | | Solicited Systemic Adverse Events<br>after first Vaccination by Diary Day<br>([Booster] Safety Analysis Set) | | Х | х |
| 27 | 3 | х | х | | | х | | | | | Solicited Systemic Adverse Events<br>after second Vaccination by Diary<br>Day ([Booster] Safety Analysis Set) | | х | х |
| 27 | 4 | х | х | | | х | | | | | Solicited Systemic Adverse Events<br>after third Vaccination by Diary Day<br>([Booster] Safety Analysis Set) | | х | х |
| 27 | 5 | | | | | х | | | | | Solicited Systemic Adverse Events<br>after Booster Vaccination by Diary<br>Day (Booster Safety Analysis Set) | | х | х |
| 28 | 1 | х | х | | | х | | | | | Greatest Diameter for Present<br>Local Reactions after each<br>Vaccination by Symptom ([Booster]<br>Safety Analysis Set) | <ul><li>Swelling</li><li>Erythema/Redness</li><li>Induration/Hardening</li></ul> | х | |


| | | | | | Ar | nalysis | | | | | Ta | able Description | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sub | | Part | Α | | | | Part B | | | | | Overall | Including |
| ID | -ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content | and by<br>age<br>cohort | statistical<br>test |
| 28 | 2 | х | х | | | х | | | | | Greatest Diameter for Present Local Reactions after first Vaccination by Symptom ([Booster] Safety Analysis Set) | | х | |
| 28 | 3 | х | х | | | х | | | | | Greatest Diameter for Present Local Reactions after second Vaccination by Symptom ([Booster] Safety Analysis Set) | | x | |
| 28 | 4 | х | х | | | х | | | | | Greatest Diameter for Present<br>Local Reactions after third<br>Vaccination by Symptom ([Booster]<br>Safety Analysis Set) | | х | |
| 28 | 5 | | | | | х | | | | | Greatest Diameter for Present Local Reactions after booster Vaccination by Symptom ([Booster] Safety Analysis Set) | | х | |
| 29 | 1 | х | х | | | х | | | | | Maximum Fever after each Vaccination ([Booster] Safety Analysis Set) | | х | |
| 29 | 2 | х | х | | | х | | | | | Maximum Fever after first<br>Vaccination ([Booster] Safety<br>Analysis Set) | | х | |
| 29 | 3 | х | х | | | х | | | | | Maximum Fever after second<br>Vaccination ([Booster] Safety<br>Analysis Set) | | х | |
| 29 | 4 | х | х | | | х | | | | | Maximum Fever after third<br>Vaccination ([Booster] Safety<br>Analysis Set) | | х | |
| 29 | 5 | | | | | х | | | | | Maximum Fever after Booster<br>Vaccination (Booster Safety<br>Analysis Set) | | х | |

| | | | | | Aı | nalysis | | | | | 1 | able Description | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sub | | Part | : <b>A</b> | | | | Part B | | | | | Overall | Including |
| ID | -ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content | and by<br>age<br>cohort | statistical<br>test |
| 30 | 1 | х | х | | | х | | | | | Number of Days with Solicited<br>Local AE by Diary Period ([Booster]<br>Safety Analysis Set) | By Symptom | х | |
| 30 | 2 | х | х | | | х | | | | | Number of Days with Solicited<br>Local AE after first Vaccination<br>([Booster] Safety Analysis Set) | By Symptom | Х | |
| 30 | 3 | х | х | | | x | | | | | Number of Days with Solicited<br>Local AE after second Vaccination<br>([Booster] Safety Analysis Set) | By Symptom | х | |
| 30 | 4 | х | х | | | х | | | | | Number of Days with Solicited<br>Local AE after third Vaccination<br>([Booster] Safety Analysis Set) | By Symptom | х | |
| 30 | 5 | | | | | х | | | | | Number of Days with Solicited<br>Local AE after Booster Vaccination<br>(Booster Safety Analysis Set) | By Symptom | х | |
| 31 | 1 | х | х | | | х | | | | | Number of Days with Solicited<br>Systemic AE by Diary Period<br>([Booster] Safety Analysis Set) | | х | |
| 31 | 2 | х | х | | | х | | | | | Number of Days with Solicited<br>Systemic AE after first Vaccination<br>([Booster] Safety Analysis Set) | | х | |
| 31 | 3 | х | х | | | х | | | | | Number of Days with Solicited<br>Systemic AE after second<br>Vaccination ([Booster] Safety<br>Analysis Set) | | х | |
| 31 | 4 | х | х | | | х | | | | | Number of Days with Solicited<br>Systemic AE after third Vaccination<br>([Booster] Safety Analysis Set) | | х | |
| 31 | 5 | | | | | х | | | | | Number of Days with Solicited<br>Systemic AE after Booster<br>Vaccination (Booster Safety<br>Analysis Set) | | х | |


| | | | | | Aı | nalysis | | | | | T | able Description | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sub | | Part | Α | | | | Part B | | | | | Overall | Including |
| ID | -ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content | and by<br>age<br>cohort | statistical<br>test |
| Unso | licited | Adverse | Events | 6 | | | | | | | | | | |
| 32 | | х | х | х | х | х | х | х | х | х | Unsolicited Adverse Events up to<br>[Time Point] by SOC and PT<br>([Booster] Safety Analysis Set) | | х | х |
| 33 | | Х | Х | X | x | х | X | х | X | х | Related Unsolicited Adverse<br>Events up to [Time Point] by SOC<br>and PT ([Booster] Safety Analysis<br>Set) | | х | x |
| 34 | | х | х | х | х | х | х | х | Х | х | Unsolicited Serious Adverse Events<br>up to [Time Point] by SOC and PT<br>([Booster] Safety Analysis Set) | | х | х |
| 35 | | х | х | х | х | х | х | х | х | х | Related Unsolicited Serious Adverse Events up to [Time Point] by SOC and PT ([Booster] Safety Analysis Set) | | х | х |
| 36 | | х | Х | х | х | х | х | х | х | х | Severe Unsolicited Adverse Events<br>up to [Time Point] by SOC and PT<br>([Booster] Safety Analysis Set) | | х | х |
| 37 | | Х | Х | х | х | х | X | х | Х | х | Related Severe Unsolicited Adverse Events up to [Time Point] by SOC and PT ([Booster] Safety Analysis Set) | | х | х |
| 38 | | х | х | х | х | х | х | х | х | х | Adverse Events of Special Interest<br>up to [Time Point] by SOC and PT<br>([Booster] Safety Analysis Set) | | х | х |
| 39 | | Х | Х | х | х | х | Х | х | х | х | Related Adverse Events of Special<br>Interest up to [Time Point] by SOC<br>and PT ([Booster] Safety Analysis<br>Set) | | х | х |
| 40 | | Х | х | Х | х | х | Х | х | Х | х | Unsolicited Adverse Events up to [Time Point] by Maximum Severity ([Booster] Safety Analysis Set) | _ | Х | х |


| | | | | | Aı | nalysis | | | | | Т | able Description | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sub | | Part | Α | | | | Part B | | | | | Overall | Including |
| ID | -ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content | and by<br>age<br>cohort | statistical<br>test |
| 41 | | Х | х | х | х | х | х | Х | х | х | Medically Attended Unsolicited<br>Adverse Events up to [Time Point]<br>by Maximum Severity ([Booster]<br>Safety Analysis Set) | | х | х |
| 42 | | Х | х | х | х | х | х | х | х | х | Adverse Events of Special Interest<br>up to [Time Point] by Maximum<br>Severity ([Booster] Safety Analysis<br>Set) | | х | х |
| 43 | | х | х | х | х | х | х | х | х | х | Unsolicited Adverse Events up to [Time Point] by Causality ([Booster] Safety Analysis Set) | | х | х |
| 44 | | Х | х | х | х | х | х | Х | Х | х | Medically Attended Unsolicited<br>Adverse Event up to [Time Point]<br>by Causality ([Booster] Safety<br>Analysis Set) | | х | х |
| 45 | | х | х | х | х | х | х | Х | х | х | Adverse Events of Special Interest<br>up to [Time Point] by Causality<br>([Booster] Safety Analysis Set) | | х | х |

### 7.1.5 Other Safety Analysis and B.b. s.l. Serostatus

| ID | | | | Ana | lysis | | | | | Table Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Part | : A | | | Pa | art B | | | | |
| | A1.1<br>A1.2 | Δ1 | A2 | A3 1 | A3.2 | ΔΔ | A5 | A6 | Α7 | Legend | Content |
| | A1.3 | / ( | / (2 | 710.1 | 710.2 | , , , | 7.0 | 7.0 | , , , | | |
| 1 | х | х | Х | х | х | Х | х | х | х | Systolic Blood Pressure [mmHg] by Visit ([Booster] Safety Analysis Set) | Including measurements after vaccinations (eCRF section "Assessment after vaccination" |
| 2 | х | Х | х | Х | х | Х | х | Х | Х | Diastolic Blood Pressure [mmHg] by Visit ([Booster] Safety Analysis Set) | See Table ID 1 |

Adapted from:
STAT03\_A Statistical Analysis Plan

without prior written consent of


| ID | | | | Ana | lysis | | | | | Table Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Part | : A | | | Pa | art B | | | | |
| | A1.1<br>A1.2 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content |
| | A1.3 | | | | | | | | | | 0 7 11 10 1 |
| 3 | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Pulse Rate [beats/min] by Visit ([Booster] Safety Analysis Set)) | See Table ID 1 |
| 4 | х | Х | Х | Х | Х | Х | Х | Х | х | Oral Body Temperature [°C] by Visit ([Booster] Safety Analysis Set) | See Table ID 1 |
| 5 | Х | х | х | Х | Х | х | х | х | х | Lyme Borreliosis Screening Results by Visit ([Booster] Safety Analysis Set) | |
| | | | | Х | | | | | | Rate of subjects who seroconverted in B.b. s.l. serostatus from Screening to Month 18/ET (Safety Analysis Set) | |
| | | | | | | | х | | | Rate of subjects who seroconverted in B.b. s.l. serostatus from Month 18 to Month 30/ET (Safety Analysis Set) | |
| 6 | | | | | | | | х | | Rate of subjects who seroconverted in B.b. s.l. serostatus from Month 30 to Month 42/ET (Safety Analysis Set) (Booster Safety Analysis Set) | |
| | | | | | | | | | Х | Seroconversion Rate of Lyme Borreliosis Screening from Visit 14 to Visit 16/ET (Booster Safety Analysis Set) | |

## 7.2 List of Data Listings

#### 7.2.1 Overall Study Information

| | | | | Ana | alysis | | | | | | Listing Description |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Par | tΑ | | | Pa | art B | | | | |
| ID | A1.1<br>A1.2<br>A1.3 | | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content |
| 1 | х | Х | х | х | х | х | х | х | х | Subject Overview | Subject ID, Age cohort, Site name, Date of signed informed consent, Planned study group, Actual study group (*), [Booster] Safety Analysis Set, Reason not in [Booster] Safety Analysis Set, [Booster] Full Analysis Set, Reason not in [Booster] Full Analysis Set, [Booster] Per-Protocol Analysis Set, Reason not in [Booster] Per-Protocol Analysis Set |

Adapted from:
STAT03\_A Statistical Analysis Plan


| | | | | Ana | alysis | | | | | | Listing Description |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Pai | rt A | | | Pa | art B | | | | |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content |
| | | | | | | | | | | | (*) Include note: Subjects are analyzed as randomized if all vaccinations were administered as planned. In case subject was mistreated at any vaccination and it can be unequivocally allocated to another study group it is analyzed in this study group. In case no unequivocally allocation can be done the subject is analyzed as "received any VLA15". |
| 2 | х | х | х | x | x | х | х | х | х | Randomization and Actual<br>Treatment Group Allocation | Subject ID, Age cohort, Randomization date, Randomization time, Randomization number, Planned treatment, Planned study group, Actual study group (*), Treatment at first vaccination, Treatment at second vaccination, Treatment at third vaccination, Treatment at booster vaccination (only applicable for Part B), |
| 3 | х | х | х | х | х | х | х | х | х | Screening Failures with Reasons | Subject ID, Age cohort, Subject withdrawal of consent, In-/exclusion criteria violated, Other reason, Specification of other reason |
| 4 | х | х | х | х | х | х | х | х | х | [Booster] In/Exclusion Criteria<br>Violations | Subject ID, Age cohort, Visit, Inclusion criterion not met / exclusion criteria met |
| 5 | х | Х | х | х | х | х | х | х | х | Study Vaccination (Vaccinated Subjects) | Subject ID, Age cohort, Planned study group, Actual study group, Visit, Vaccination administered, Reason vaccination not administered, Vaccination date, Vaccination time, Kit number, Location, Other location (specification/reason) |
| 6 | х | Х | х | х | х | х | х | х | х | Visit Log (Vaccinated Subjects) | Subject ID, Age cohort, Planned s group, Actual study group, Visit, Visit performed, Visit date, Reason visit not performed, Type of contact, Outside time window, Deviation from time window [days], Reason outside time window, Age at date of visit [years], Gender, Menarche onset, Continue with booster phase (A.3.2-A.7 only), Visit V8B performed on the same day as visit V8 (A.3.2-A.7 only), Reason for unscheduled visit |
| 7 | х | Х | х | х | х | х | х | х | х | Visits Performed as Phone Call<br>(Vaccinated Subjects) | Subject ID, Age cohort, Planned study group, Actual study group, Visit, Visit performed (phone/video call), Visit date, Outside time window, Deviation from time window [days], Reason outside time window, Age at visit date, Immunogenicity blood sample collected |
| 8 | х | х | х | Х | х | Х | Х | Х | Х | Missed Visits, Missed<br>Vaccinations, Early Terminations | Subject ID, Age cohort, Planned study group, Actual study group, Visit attendance status of subject, All vaccinations administered, |

| | Analysis Part A Part B | | | | | | | | | | Listing Description |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Pa | rt A | | | Pa | art B | } | | | |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content |
| | | | | | | | | | | up to [Time Point]: Part I<br>(Vaccinated Subjects) | Primary reason treatment discontinuation, Other reason treatment discontinuation, AE leading to treatment discontinuation, Reason for recommended withdrawal for treatment discontinuation, Individual stopping criteria fulfilled, AE Term (stopping criteria) |
| 9 | Х | х | х | Х | Х | х | x | х | х | Missed Visits, Missed<br>Vaccinations, Early Terminations<br>up to [Time Point]: Part II<br>(Vaccinated Subjects) | Subject ID, Age cohort, Planned study group, Actual study group, Primary reason same for IMP disc. and ET, Primary reason for early termination Other reason for early termination, AE leading to early termination, Reason for recommended withdrawal (early termination), Death date, Primary cause of death, Date of study discontinuation (ET), Last attended scheduled visit before ET |
| 10 | х | х | х | х | х | х | х | х | х | Relevant and Non-relevant<br>Protocol Deviations (Vaccinated<br>Subjects) | Subject ID, Age cohort, Planned study group, Actual study group, Visit, PD category, PD Description, Classification (PPAS), Reason for classification (PPAS), Related to COVID-19 pandemic, |
| 11 | х | х | х | х | х | х | х | х | х | Major and minor Protocol<br>Deviations (Vaccinated Subjects) | Subject ID, Age cohort, Planned study group, Actual study group, Visit, PD category, PD Description, Classification by CRA, Related to COVID-19 pandemic |

#### 7.2.2 Baseline Evaluation

| | | | | Ana | lysis | | | | | Li | isting Description |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Part | ŧΑ | , | | Pa | art B | | , | | |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content |
| 1 | x | x | x | x | x | x | x | x | x | Demographic Information (Vaccinated Subjects) | Subject ID, Planned study group, Actual study group (*), Received any VLA15 vaccination, Year of birth, Age at screening [years], Age cohort, Gender, Females with childbearing potential, Reason non-childbearing potential (incl. specification of other reason), Race, (incl. specification of other race), Ethnicity, Body height [cm], Body weight [kg] at, BMI [kg/m2] "not done" will be displayed in column for body height or body weight in case "not done" is ticked in the eCRF for the respective measurement. (*) Include note: Subjects are analyzed as randomized if all vaccinations were administered as planned. In case subject was mistreated at any vaccination and it can be unequivocally allocated to another study group it is analyzed in this study group. In case no unequivocally allocation can be done the subject is analyzed as "received any VLA15". |
| 2 | x | х | х | х | х | х | х | х | х | Physical Examination (Vaccinated Subjects) | Subject ID, Age cohort, Planned study group, Actual study group, Physical examination performed, Reason physical examination not performed, Examination date |
| 3 | Х | х | х | х | х | х | х | х | х | ECG (Vaccinated Subjects) | Subject ID, Age cohort, Planned study group, Actual study group, ECG performed, Reason ECG not performed, ECG date, ECG result, Clinically relevant |
| 4 | Х | х | х | х | х | х | х | х | х | HIV Test (Vaccinated Subjects) | Subject ID, Age cohort, Planned study group, Actual study group, HIV test performed, Reason test not performed, Date test performed, Result |
| 5 | Х | Х | Х | х | х | х | Х | х | Х | Medical History (Vaccinated Subjects) | Subject ID, Age cohort, Planned study group, Actual study group, Condition, MedDRA SOC [Version], MedDRA |

Adapted from:
STAT03\_A Statistical Analysis Plan
Confidential and intellectual property of without prior written consent of


| | | | | Ana | lysis | | | | | Li | isting Description |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Part | tΑ | | | Pa | art B | | | | |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content |
| | | | | | | | | | | | PT [Version], Start Date, End Date, Ongoing at study entry, Ongoing at Day 1 |
| 6 | Х | х | х | х | х | х | х | х | х | Prior Medications (Vaccinated Subjects) | Subject ID, Age cohort, Planned study group, Actual study group, Medication or therapy, Start date, End date, ATC term level 2 [Version], ATC term level 3 [version], Dose, Dose Unit (incl. specification other), Dose Form (incl. specification other), Dose frequency (incl. specification other), Dose route (incl. specification other), Indication category, Indication |
| 7 | х | х | х | х | х | х | х | х | х | Concomitant Medications started up to [Time Point] (Vaccinated Subjects) | See Content ID 6 |
| 8 | х | х | х | х | х | х | х | х | х | Prior Procedures (Vaccinated Subjects) | Subject ID, Age cohort, Planned study group, Actual study group, Procedure, MedDRA SOC [Version], MedDRA PT [Version], Start date, Ongoing at study end, End date, Indication category, Indication |
| 9 | х | х | х | х | х | х | х | х | х | Concomitant Procedures started up to [Time Point] (Vaccinated Subjects) | see Content ID 8 |
| 10 | х | х | х | x | х | х | х | х | х | Vaccination History (Vaccinated Subjects) | Subject ID, Age cohort, Planned study group, Actual study group, Vaccination date, Vaccination (indication or trade name), ATC term level 3 [Version] |

# 7.2.3 Immunogenicity Analysis

| ID | | | | Ana | lysis | | | | | Listing Descrip | tion |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Part | : A | | | Pa | art B | | | | |
| | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | Α7 | Legend | Content |
| 1 | х | х | x | x | х | x | х | х | х | ELISA Immunogenicity Results (Vaccinated Subjects) | Subject ID, Age cohort, Planned study group, Per-protocol Analysis Set, Visit, Visit date, Visit time, Sample collected, Reason for not collected, Sample included in PP analysis, Sample ID, Plate ID, Serotype, ELISA IgG titer [U/mL] (measured), ELISA IgG titer [U/mL] (analysis), Sample status, Fold increase from baseline, Seroconversion from baseline |
| 2 | Х | х | х | х | Х | х | х | х | х | ELISA Immunogenicity Results for Combined Serotypes (Vaccinated Subjects) | Subject number, Age cohort, Planned study group, Per-protocol Analysis Set, Sample included in PP analysis, Visit, Visit date, Visit time, Seroconversion for all six serotypes ST1-6 from baseline, Seroconversion for ST1 and ST2 from baseline |
| • | | | | | • | • | | | | CCI | |
| | | | | | • | • | | | | | |

Adapted from:
STAT03\_A Statistical Analysis Plan
Confidential and intellectual property of without prior written consent of


#### 7.2.4 Adverse Events

| | | | | Aı | nalysis | | | | | Listing | Description |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Part | : A | | | | Part B | | | | |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content |
| Solicit | ted and l | Jnsolio | cited A | dverse | Events | 3 | | | | | |
| 1 | х | х | х | x | x | x | x | х | х | Serious Adverse Events up to [Time Point] (solicited and unsolicited) - Part I (Vaccinated Subjects) | Subject ID, Age cohort, Actual study group (*), Record ID, Solicited/unsolicited, Adverse event, MedDRA SOC [Version], MedDRA PT [Version], Severity, Serious, SAE criteria, SAE onset date, Event considered as AESI, Medically attended, Causality (*) Include note: Subjects are analyzed as randomized if all vaccinations were administered as planned. In case subject was mistreated at any vaccination and it can be unequivocally allocated to another study group it is analyzed in this study group. In case no unequivocally allocation can be done the subject is analyzed as "received any VLA15". |
| 2 | х | Х | Х | X | Х | Х | х | х | X | Serious Adverse Events up to [Time Point] (solicited and unsolicited) – Part II (Vaccinated Subjects) | Subject ID, Age cohort, Actual study group (*), Record ID, solicited/unsolicited, Adverse event, Action taken on IMP, Other action taken, Outcome, Start date, Start time, Study day of onset, Onset after vaccination, Onset (relative to that vaccination) [days], Treatment received at this vaccination,, End date/ongoing at final examination, End time, Estimated duration of AE (incl. missing stop date) [days] See content ID 1 |
| 3 | х | Х | х | х | Х | х | х | Х | х | Medically Attended Adverse Events up<br>to [Time Point] (solicited and<br>unsolicited) – Part I (Vaccinated<br>Subjects) | See content ID 1 |

Adapted from:
STAT03\_A Statistical Analysis Plan


| | | | | Α | nalysis | | | | | Listing | Description |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Part | t A | | | | Part B | | | | |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content |
| 4 | х | х | Х | х | х | Х | Х | Х | х | Medically Attended Adverse Events<br>(solicited and unsolicited) – Part II<br>(Vaccinated Subjects) | See content ID 2 |
| 5 | х | х | х | х | х | х | х | х | х | Adverse Events Resulting in Death (solicited and unsolicited) – Part I (Vaccinated Subjects) | See content ID 1 |
| 6 | х | х | х | х | х | х | х | х | х | Adverse Events Resulting in Death (solicited and unsolicited) – Part II (Vaccinated Subjects) | See content ID 2 |
| 7 | x | х | х | х | х | х | х | х | х | Adverse Events with Missing Assessment (eCRF Section "AE log") – Part I (Vaccinated Subjects) | See content ID 1 |
| 8 | x | х | х | х | х | х | х | х | х | Adverse Events with Missing Assessment (eCRF Section "AE log") – Part II (Vaccinated Subjects) | See content ID 2 |
| Unsol | icited Ad | verse | Events | 5 | | | | | | | |
| 9 | X | Х | х | х | Х | Х | Х | Х | х | Unsolicited Adverse Events up to [Time Point] – Part I (Vaccinated Subjects) | Subject ID, Age cohort, Actual study group (*), Record ID, Adverse event, MedDRA SOC [Version], MedDRA PT [Version], Severity, Serious, SAE criteria, SAE onset date, Event considered as AESI, Medically attended, Causality |
| 10 | x | X | х | x | x | X | х | X | х | Unsolicited Adverse Events up to [Time Point] - Part II (Vaccinated Subjects) | Subject ID, Age cohort, Actual study group (*), Record ID, Adverse event, Action taken on IMP, Other action taken, Outcome, Start date, Start time, Study day of onset, Onset after vaccination Onset (relative to previous vaccination) [days], Treatment received at this vaccination, End date/ongoing at final examination, Estimated duration of AE (incl. missing stop date) [days] |

| | | | | Α | nalysis | | | | | Listing | Description |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Parl | t A | | | | Part B | | | | |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content |
| 11 | х | х | х | х | х | х | х | х | х | Related Unsolicited Adverse Events up<br>to [Time Point] – Part I (Vaccinated<br>Subjects) | See content ID 9 |
| 12 | х | х | x | х | х | х | х | х | х | Related Unsolicited Adverse Events up<br>to [Time Point] – Part II (Vaccinated<br>Subjects) | See content ID 10 |
| 13 | x | X | х | Х | x | X | х | х | х | Related Unsolicited Adverse Events up to [Time Point] per SOC (Vaccinated Subjects) | Subject ID, Actual study group (*), Age cohort, Adverse Event, MedDRA SOC [Version], MedDRA PT [Version], Onset after vaccination, Onset (relative to previous vaccination) [days], Treatment received at this vaccination, Estimated duration of AE (incl. missing stop date) [days], Severity Listing will be presented by SOC, Age Cohort, and Subject ID. |
| 14 | х | х | х | х | х | х | х | х | х | Severe Unsolicited Adverse Events up<br>to [Time Point] – Part I (Vaccinated<br>Subjects) | See content ID 9 |
| 15 | х | х | х | х | х | х | х | х | х | Severe Unsolicited Adverse Events up<br>to [Time Point] – Part II (Vaccinated<br>Subjects) | See content ID 10 |
| 16 | х | x | x | х | х | x | х | x | х | Unsolicited Adverse Events Leading to Withdrawal from Further Vaccination – Part I (Vaccinated Subjects) | See content ID 9 |
| 17 | Х | Х | х | х | х | Х | х | х | х | Unsolicited Adverse Events Leading to<br>Withdrawal from Further Vaccination –<br>Part II (Vaccinated Subjects) | See content ID 10 |
| 18 | Х | Х | х | х | х | Х | х | Х | х | Unsolicited Adverse Events Leading to<br>Withdrawal from the Study – Part I<br>(Vaccinated Subjects) | See content ID 9 |

| | | | | Aı | nalysis | | | | | Listing | Description |
|---|---|---|---|---|---|---|---|---|---|---|---|
| ID | A1.1<br>A1.2<br>A1.3 | Part<br>A1 | A2 | A3.1 | A3.2 | A4 | Part B<br>A5 | A6 | A7 | Legend | Content |
| 19 | X X | Х | Х | х | х | Х | Х | Х | Х | Unsolicited Adverse Events Leading to<br>Withdrawal from the Study – Part II<br>(Vaccinated Subjects) | See content ID 10 |
| 20 | х | х | х | х | х | х | х | х | х | Adverse Events of Special Interest –<br>Part I (Vaccinated Subjects) | See content ID 9 |
| 21 | х | х | х | х | х | х | х | х | х | Adverse Events of Special Interest –<br>Part II (Vaccinated Subjects) | See content ID 10 |
| Solicit | ed Adve | rse Ev | ents | | | | | | | | |
| 22 | х | х | | | х | | | | | Solicited Adverse Events Entered in<br>eCRF Section "AE log") – Part I<br>(Vaccinated Subjects) | See content ID 9 |
| 23 | х | х | | | х | | | | | Solicited Adverse Events Entered in<br>eCRF Section "AE log") – Part II<br>(Vaccinated Subjects) | See content ID 10 |
| 24 | х | х | | | х | | | | | Solicited Adverse Events - Assessment<br>After Vaccination (Vaccinated Subjects) | Subject ID, Age cohort, Actual study group, Visit, Diameter [cm], Oral body temperature [°C], Grading (Investigator's assessment), Any medication taken, Symptom fulfilling any SAE criteria Only symptoms with "Symptom present" = |
| | | | | | | | | | | Calinited Advarsa Events (Investigator | "yes" in eCRF are displayed |
| 25 | х | х | | | х | | | | | Solicited Adverse Events – (Investigator Assessment, Vaccinated Subjects) | Subject ID, Age cohort, Actual study group, Symptom, Vaccination period, Treatment received at this vaccination, Symptom present, Severity (Investigator), Symptom medically attended, Medication taken/received due to this symptom, Max. diameter [cm], Symptom fulfilling any SAE criteria, Withdrawn from further IMP due to |

| | | | | Aı | nalysis | | | | | Listing | Description |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Part | tΑ | | | | Part B | | | | |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content |
| | | | | | | | | | | | symptom, Withdrawn from study due to symptom |
| | | | | | | | | | | | Based on only symptoms with "Symptom present" = "yes" in eCRF are displayed |
| 26 | x | х | | | x | | | | | Solicited Adverse Events by Diary Day –<br>Part I (Subjects eDiary, Vaccinated<br>Subjects) | Subject ID, Age cohort, Actual study group, Symptom, Diary time point, Treatment received at this vaccination, Severity of symptom, Needed to take medicine due to symptom, Specification of taken medication(s), Needed to see a doctor due to symptom, Specification of care given for symptom, Symptom end date, Symptom ongoing beyond Day 6 after vaccination,, Max. diameter (cm), Oral body temperature [°C], Diameter/Temperature not measured Based on only symptoms with "Symptom present" = "yes" in eCRF are displayed |
| 27 | х | Х | | | X | | | | | Solicited Adverse Events by Diary Day –<br>Part II (Subjects eDiary, Vaccinated<br>Subjects) | Subject ID, Age cohort, Actual study group, Symptom, Diary time point, Treatment received at this vaccination, Date temperature measurement, Time temperature measurement, Additional measurement(s) of body temperature, Specification of other comment Based on only symptoms with "Symptom present" = "yes" in eCRF are displayed |
| 28 | х | Х | х | | х | х | х | Х | х | Body Temperature in Case of Fever (Vaccinated Subjects) | Subject ID, Age cohort, Actual study group, Diary time point, Treatment received at this vaccination, Date of measurement, Time of measurement, Oral body temperature [°C] |

Adapted from: STATO3\_A Statistical Analysis Plan Version 6.0, Effective Date 16-Feb-2018

without prior written consent of


| | | | | Aı | nalysis | | | | | Listing | Description |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Part | : A | | | | Part B | , | | | |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content |
| 29 | х | х | | | х | | | | | Additional Temperature Measurements (Subjects eDiary, Vaccinated Subjects) | Subject ID, Age cohort, Actual study group, Date of measurement, Time of measurement, Oral body temperature [°C] |
| 30 | х | х | | | х | | | | | Other Symptoms (Subjects eDiary, - Vaccinated Subjects) | Subject ID, Age cohort, Actual study group, Symptom, Date symptom started, Date symptom ended, Medical advice seemed, Severity of the symptom, Comment |
| 31 | х | х | | | х | | | | | Severe Solicited Adverse Events -<br>Assessment After Vaccination<br>(Vaccinated Subjects) | See content ID 24 |
| 32 | х | х | | | х | | | | | Severe Solicited Adverse Events<br>(Investigator Assessment, Vaccinated<br>Subjects) | See content ID 25 |
| 33 | х | х | | | х | | | | | Severe Solicited Adverse Events by<br>Diary Day – Part I (Subjects eDiary,<br>Vaccinated Subjects) | See content ID 26 |
| 34 | х | х | | | х | | | | | Severe Solicited Adverse Events by<br>Diary Day – Part II (Subjects eDiary,<br>Vaccinated Subjects) | See content ID 27 |
| 35 | х | х | | | х | | | | | Solicited Adverse Events Leading to<br>Withdrawal From Further Vaccination<br>(Investigator Assessment, Vaccinated<br>Subjects) | See content ID 24 |
| 36 | х | х | | | х | | | | | Solicited Adverse Events Leading to<br>Withdrawal From Study (Investigator<br>Assessment, Vaccinated Subjects) | See content ID 25 |
| 37 | х | х | | | х | | | | | Solicited Adverse With Missing<br>Assessments (Investigator Assessment,<br>Vaccinated Subjects) | See content ID 25 |
| 38 | Х | Х | | | х | | | | | Solicited Adverse With Missing Assessments by Diary Day – Part I (Subjects eDiary, Vaccinated Subjects) | See content ID 26 |


| | | | | Aı | nalysis | | | | | Listing | Description |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Part A Part B | | | | | | | | | | |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content |
| 39 | х | х | | | х | | | | | Solicited Adverse With Missing Assessments by Diary Day – Part II (Subjects eDiary, Vaccinated Subjects) | See content ID 27 |

### 7.2.5 Other Safety Analysis and B.b. s.l. Serostatus

| | | | | An | alysis | | | | | Lis | sting Description |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Pa | rt A | | | Pa | art B | } | | | |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content |
| 1 | х | х | | | х | | | | | Assessment After Vaccination Performed (Vaccinated Subjects) | Subject ID, Age cohort, Actual study group, Visit, Observation performed, Reason observation not performed, Any solicited event during observation Physical examination and vital sign information will be listed in the respective Listing below |
| 2 | x | х | х | x | х | x | х | x | х | Vital Signs [Including Assessment After<br>Vaccination Results] (Vaccinated Subjects) | Subject ID, Age cohort, Actual study group, Visit (incl. specifier), Vital signs collected, Reason vital signs not collected, Collection date, Collection time, Systolic blood pressure [mmHg], Systolic blood pressure clinically relevant, Diastolic blood pressure [mmHg], Diastolic blood pressure clinically relevant, Pulse rate [beats/min], Pulse rate clinically relevant, Oral body temperature [°C], Oral boy temperature clinically relevant |
| 3 | х | х | х | х | х | х | х | х | х | Physical Examination [Including<br>Assessment After Vaccination Results]<br>(Vaccinated Subjects) | Subject ID, Age cohort, Actual study group, Visit (incl. specifier), Examination date, Examination time, Category, Physical examination performed, Reason physical examination/observation not performed |
| 4 | х | х | х | х | х | Х | х | х | х | Pregnancy Test (Vaccinated Female Subjects) | Subject ID, Age cohort, Actual study group, Visit, Pregnancy test date, Pregnancy test time, Pregnancy |

| | | | | Ana | alysis | | | | | Lis | ting Description |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Pai | rt A | | | Pa | art B | | | | |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | Content |
| | | | | | | | | | | | test performed, Reason pregnancy test not performed, Pregnancy test type, Pregnancy test result |
| 5 | х | х | х | х | х | х | х | х | х | Injection Site Inspection (Vaccinated Subjects) | Subject ID, Age cohort, Actual study group, Visit, Inspection date, Inspection time, linjection site inspected, Reason inspection not performed, Any findings |
| 6 | Х | х | | | Х | | | | | Vaccination Delay Criteria (Vaccinated Subjects) | Subject ID, Age cohort, Actual study group, Visit,<br>Checklist question, Answer |
| 7 | х | х | | | | | х | х | х | Lyme Borreliosis Screening (Vaccinated Subjects) | Subject ID, Age cohort, Actual study group, Visit, Collection date, Sample collected, Reason not collected, Borrelia burgdorferi s.l. IgG (Diasorin), Borrelia burgdorferi s.l. IgM (Diasorin), Borrelia IgG antibodies (Virachip), Borrelia IgM antibodies (Virachip), Interp. B.b. s.l. serostatus (derived) |

#### List of Figures 7.3

### 7.3.1 Immunogenicity Analysis

| | | | | Ar | alysis | | | | | Figure Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Part A Part B | | | | | | | | | | |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4<br>3 | A5 | A6 | A7 | Legend | by age<br>cohort <sup>5</sup> |
| 1 | х | Х | Х | Х | Х | х | х | х | Х | Bar Chart: ELISA OspA Specific IgG Antibodies (GMT) at Day 85 by OspA Specific Serotype and Study Group ([Booster] Per-Protocol Analysis Set) | х |

STATO3\_A Statistical Analysis Plan Version 6.0, Effective Date 16-Feb-2018 without prior written consent of

<sup>&</sup>lt;sup>5</sup> Detailed layout of the figures will be discussed during the review of the dummy analysis (see Section 8). Figures stratified by age cohort might be presented in separate plots. Adapted from:

| | Analysis | | | | | | | | | Figure Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Part | Α | | | | Part B | } | | | Overall and |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4<br>3 | A5 | A6 | A7 | Legend | by age<br>cohort <sup>5</sup> |
| 2 | х | х | х | Х | Х | х | х | Х | Х | Bar Chart: ELISA OspA Specific IgG Antibodies (GMT) at Day 180 by OspA Specific Serotype and Study Group ([Booster] Per-Protocol Analysis Set) | х |
| 3 | х | Х | х | Х | х | Х | х | х | Х | Bar Chart: ELISA OspA Specific IgG Antibodies (GMT) at Day 194 by OspA Specific Serotype and Study Group ([Booster] Per-Protocol Analysis Set) | х |
| 4 | х | Х | х | Х | х | Х | х | х | Х | Bar Chart: ELISA OspA Specific IgG Antibodies (GMT) at Day 208 by OspA Specific Serotype and Study Group ([Booster] Per-Protocol Analysis Set) | х |
| 5 | | | х | Х | Х | х | х | х | Х | Bar Chart: ELISA OspA Specific IgG Antibodies (GMT) at Day 365 by OspA Specific Serotype and Study Group ([Booster]Per-Protocol Analysis Set) | х |
| 6 | | | | Х | х | х | х | х | Х | Bar Chart: ELISA OspA Specific IgG Antibodies (GMT) at Month 18 by OspA Specific Serotype and Study Group ([Booster]Per-Protocol Analysis Set) | х |
| 7 | | | | | Х | Х | х | Х | Х | Bar Chart: ELISA OspA Specific IgG Antibodies (GMT) at Month 19 by OspA Specific Serotype and Study Group (Booster Per-Protocol Analysis Set) | х |
| 8 | | | | | | х | х | Х | Х | Bar Chart: ELISA OspA Specific IgG Antibodies (GMT) at Month 23 by OspA Specific Serotype and Study Group (Booster Per-Protocol Analysis Set) | х |
| 9 | | | | | | х | х | Х | Х | Bar Chart: ELISA OspA Specific IgG Antibodies (GMT) at Month 26 by OspA Specific Serotype and Study Group (Booster Per-Protocol Analysis Set) | х |
| 10 | | | | | | | х | Х | Х | Bar Chart: ELISA OspA Specific IgG Antibodies (GMT) at Month 30 by OspA Specific Serotype and Study Group (Booster Per-Protocol Analysis Set) | х |
| 11 | | | | | | | | Х | Х | Bar Chart: ELISA OspA Specific IgG Antibodies (GMT) at Month 36 by OspA Specific Serotype and Study Group (Booster Per-Protocol Analysis Set) | х |
| 12 | | | | | | | | Х | Х | Bar Chart: ELISA OspA Specific IgG Antibodies (GMT) at Month 42 by OspA Specific Serotype and Study Group (Booster Per-Protocol Analysis Set) | х |
| 13 | | | | | | | | | Х | Bar Chart: ELISA OspA Specific IgG Antibodies (GMT) at Month 48 by OspA Specific Serotype and Study Group (Booster Per-Protocol Analysis Set) | х |
| 14 | | | | | | | | | Х | Bar Chart: ELISA OspA Specific IgG Antibodies (GMT) at Month 54 by OspA Specific Serotype and Study Group (Booster Per-Protocol Analysis Set) | х |
| 15 | х | Х | Х | Х | х | х | х | Х | Х | Bar Chart: ELISA OspA Specific IgG Antibodies (GMT) Over Time in Study Group 1 by OspA Specific Serotype ([Booster] Per-Protocol Analysis Set) | х |
| 16 | х | Х | Х | Х | х | х | х | Х | Х | Bar Chart: ELISA OspA Specific IgG Antibodies (GMT) Over time in Study Group 2 by OspA Specific Serotype ([Booster] Per-Protocol Analysis Set) | х |
| 17 | Х | х | х | х | х | х | х | Х | х | Bar Chart: ELISA OspA Specific IgG Antibodies (GMT) at Day 208 in Study Group 1 by OspA Specific Serotype and Age Cohort ([Booster] Per-Protocol Analysis) | х |


| | Analysis | | | | | | | | | Figure Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Part | Α | | | | Part B | | | | Overall and |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4<br>3 | A5 | A6 | A7 | Legend | by age<br>cohort <sup>5</sup> |
| 18 | х | Х | Х | Х | Х | Х | х | Х | Х | Bar Chart: ELISA OspA Specific IgG Antibodies (GMT) at Day 208 in Study Group 2 by OspA Specific Serotype and Age Cohort ([Booster] Per-Protocol Analysis) | х |
| 19 | | | | | Х | Х | х | Х | Х | Bar Chart: ELISA OspA Specific IgG Antibodies (GMT) at Month 19 in Study Group 1 by OspA Specific Serotype and Age Cohort (Booster Per-Protocol Analysis) | х |
| 20 | | | | | Х | Х | х | Х | Х | Bar Chart: ELISA OspA Specific IgG Antibodies (GMT) at Month 19 in Study Group 2 by OspA Specific Serotype and Age Cohort ([Booster] Per-Protocol Analysis) | х |
| 21 | х | Х | Х | Х | Х | Х | х | Х | Х | Bar Chart: ELISA Seroconversion Rate at Day 85 by OspA Specific Serotype and Study Group ([Booster] Per-Protocol Analysis Set) | х |
| 22 | х | х | х | Х | х | х | х | Х | Х | Bar Chart: ELISA Seroconversion Rate at Day 180 by OspA Specific Serotype and Study Group ([Booster] Per-Protocol Analysis Set) | х |
| 23 | х | Х | Х | Х | Х | Х | х | Х | Х | Bar Chart: ELISA Seroconversion Rate at Day 194 by OspA Specific Serotype and Study Group ([Booster] Per-Protocol Analysis Set) | х |
| 24 | х | Х | Х | Х | Х | Х | х | Х | Х | Bar Chart: ELISA Seroconversion Rate at Day 208 by OspA Specific Serotype and Study Group ([Booster] Per-Protocol Analysis Set) | х |
| 25 | | | х | Х | х | х | х | Х | Х | Bar Chart: ELISA Seroconversion Rate at Day 365 by OspA Specific Serotype and Study Group ([Booster] Per-Protocol Analysis Set) | х |
| 26 | | | | Х | Х | Х | х | Х | Х | Bar Chart: ELISA Seroconversion Rate at Month 18 by OspA Specific Serotype and Study Group ([Booster] Per-Protocol Analysis Set) | х |
| 27 | | | | | Х | х | х | Х | Х | Bar Chart: ELISA Seroconversion Rate at Month 19 by OspA Specific Serotype and Study Group (Booster Per-Protocol Analysis Set) | х |
| 28 | | | | | | Х | х | Х | Х | Bar Chart: ELISA Seroconversion Rate at Month 23 by OspA Specific Serotype and Study Group (Booster Per-Protocol Analysis Set) | х |
| 29 | | | | | | Х | х | Х | Х | Bar Chart: ELISA Seroconversion Rate at Month 26 by OspA Specific Serotype and Study Group (Booster Per-Protocol Analysis Set) | х |
| 30 | | | | | | | х | Х | Х | Bar Chart: ELISA Seroconversion Rate at Month 30 by OspA Specific Serotype and Study Group (Booster Per-Protocol Analysis Set) | х |
| 31 | | | | | | | | Х | х | Bar Chart: ELISA Seroconversion Rate at Month 36 by OspA Specific Serotype and Study Group at ([Booster] Per-Protocol Analysis Set) | х |
| 32 | | | | | | | | Х | Х | Bar Chart: ELISA Seroconversion Rate at Month 42 by OspA Serotype and Study Group ([Booster] Per-Protocol Analysis Set) | х |
| 33 | | | | | | | | | х | Bar Chart: ELISA Seroconversion Rate at Month 48 by OspA Specific Serotype and Study Group ([Booster] Per-Protocol Analysis Set) | х |


| | | | | Ar | nalysis | | | | | Figure Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Part | Α | , | | | Part B | 3 | , | | Overall and |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4<br>3 | A5 | A6 | A7 | Legend | by age<br>cohort <sup>5</sup> |
| 34 | | | | | | | | | Х | Bar Chart: ELISA Seroconversion Rate at Month 54 by OspA Specific Serotype and Study Group ([Booster] Per-Protocol Analysis Set) | Х |
| 35 | х | Х | Х | Х | Х | х | х | Х | Х | Bar Chart: ELISA Seroconversion Rate for OspA STs 1-6 Combined Over Time vs. Study Group ([Booster] Per-Protocol Analysis Set) | Х |
| 36 | х | Х | Х | Х | Х | х | х | х | Х | Bar Chart: ELISA Seroconversion Rate for OspA Serotypes ST1 and ST2<br>Combined Over Time vs. Study Group ([Booster] Per-Protocol Analysis Set) | х |
| 37 | х | х | х | Х | Х | х | х | х | Х | Line Chart: ELISA OspA Specific IgG Antibodies (GMT) Over Time vs. Study Group for ST1 ([Booster] Per-Protocol Analysis Set) | х |
| 38 | х | х | х | х | х | х | х | х | Х | Line Chart: ELISA OspA Specific IgG Antibodies (GMT) Over Time vs. Study Group for ST2 ([Booster] Per-Protocol Analysis Set) | х |
| 39 | х | х | х | х | х | х | х | Х | Х | Line Chart: ELISA OspA Specific IgG Antibodies (GMT) Over Time vs. Study Group for ST3 ([Booster] Per-Protocol Analysis Set) | х |
| 40 | х | Х | Х | Х | Х | х | х | Х | Х | Line Chart: ELISA OspA Specific IgG Antibodies (GMT) Over Time vs. Study Group for ST4 ([Booster] Per-Protocol Analysis Set) | х |
| 41 | х | Х | Х | Х | Х | х | х | Х | Х | Line Chart: ELISA OspA Specific IgG Antibodies (GMT) Over Time vs. Study Group for ST5 ([Booster] Per-Protocol Analysis Set) | Х |
| 42 | х | Х | х | Х | Х | х | х | Х | Х | Line Chart: ELISA OspA Specific IgG Antibodies (GMT) Over Time vs. Study Group for ST6 ([Booster] Per-Protocol Analysis Set) | х |
| 43 | х | Х | Х | Х | Х | х | х | Х | Х | Line Chart: ELISA OspA Specific IgG Antibodies (GMT) Over Time in Study Group 1 by OspA Specific Serotype ([Booster] Per-Protocol Analysis Set) | х |
| 44 | х | Х | Х | Х | Х | х | х | Х | Х | Line Chart: ELISA OspA Specific IgG Antibodies (GMT) Over Time in Study Group 2 by OspA Specific Serotype ([Booster] Per-Protocol Analysis Set) | Х |
| 45 | х | Х | х | х | х | х | х | Х | х | Reverse Cumulative Distribution Curves for ELISA Study Group 1: Percentage of Subjects vs. OspA ST1 Specific IgG Titer (GMT) by Visit ([Booster] Per-Protocol Analysis Set) | х |
| 46 | Х | х | х | Х | Х | х | х | Х | х | Reverse Cumulative Distribution Curves for ELISA Study Group 2: Percentage of Subjects vs. OspA ST1 Specific IgG Titer (GMT) by Visit ([Booster] Per-Protocol Analysis Set) | х |
| 47 | Х | х | х | Х | Х | х | Х | Х | х | Reverse Cumulative Distribution Curves for ELISA Study Group 1: Percentage of Subjects vs. OspA ST2 Specific IgG Titer (GMT) by Visit ([Booster] Per-Protocol Analysis Set) | Х |

| | Analysis | | | | | | | | | Figure Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Part | Α | r | | | Part E | } | 1 | | Overall and |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4<br>3 | A5 | A6 | A7 | Legend | by age<br>cohort <sup>5</sup> |
| 48 | х | х | х | х | х | х | х | Х | х | Reverse Cumulative Distribution Curves for ELISA Study Group 2: Percentage of Subjects vs. OspA ST2 Specific IgG Titer (GMT) by Visit ([Booster] Per-Protocol Analysis Set) | х |
| 49 | х | х | х | х | х | х | х | Х | х | Reverse Cumulative Distribution Curves for ELISA Study Group 1: Percentage of Subjects vs. OspA ST3 Specific IgG Titer (GMT) by Visit ([Booster] Per-Protocol Analysis Set) | Х |
| 50 | х | х | Х | х | х | х | х | Х | х | Reverse Cumulative Distribution Curves for ELISA Study Group 2: Percentage of Subjects vs. OspA ST3 Specific IgG Titer (GMT) by Visit ([Booster] Per-Protocol Analysis Set) | х |
| 51 | х | х | Х | х | х | х | Х | Х | х | Reverse Cumulative Distribution Curves for ELISA Study Group 1: Percentage of Subjects vs. OspA ST4 Specific IgG Titer (GMT) by Visit ([Booster] Per-Protocol Analysis Set) | х |
| 52 | х | х | Х | х | х | х | х | Х | х | Reverse Cumulative Distribution Curves for ELISA Study Group 2: Percentage of Subjects vs. OspA ST4 Specific IgG Titer (GMT) by Visit ([Booster] Per-Protocol Analysis Set) | х |
| 53 | х | х | Х | х | х | х | х | Х | х | Reverse Cumulative Distribution Curves for ELISA Study Group 1: Percentage of Subjects vs. OspA ST5 Specific IgG Titer (GMT) by Visit ([Booster] Per-Protocol Analysis Set) | х |
| 54 | х | х | Х | х | х | х | Х | Х | Х | Reverse Cumulative Distribution Curves for ELISA Study Group 2: Percentage of Subjects vs. OspA ST5 Specific IgG Titer (GMT) by Visit ([Booster] Per-Protocol Analysis Set) | х |
| 55 | х | х | Х | х | х | х | х | Х | х | Reverse Cumulative Distribution Curves for ELISA Study Group 1: Percentage of Subjects vs. OspA ST6 Specific IgG Titer (GMT) by Visit ([Booster] Per-Protocol Analysis Set) | х |
| 56 | Х | х | х | х | х | х | Х | Х | х | Reverse Cumulative Distribution Curves for ELISA Study Group 2: Percentage of Subjects vs. OspA ST6 Specific IgG Titer (GMT) by Visit ([Booster] Per-Protocol Analysis Set) | х |
| 57 | Х | х | х | Х | Х | х | Х | Х | х | Reverse Cumulative Distribution Curves at Day 208 for ELISA Study Group 1 and 2: Percentage of Subjects vs. OspA ST1 Specific IgG Titer (GMT) by Age Cohort ([Booster] Per-Protocol Analysis Set) | |

| | | | | Ar | nalysis | | | | | Figure Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Part | Α | | | | Part E | 3 | | | Overall and |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | <b>A4</b> 3 | A5 | A6 | A7 | Legend | by age<br>cohort <sup>5</sup> |
| 58 | х | х | Х | х | х | х | Х | Х | х | Reverse Cumulative Distribution Curves at Day 208 for ELISA Study Group 1 and 2: Percentage of Subjects vs. OspA ST2 Specific IgG Titer (GMT) by Age Cohort ([Booster] Per-Protocol Analysis Set) | |
| 59 | х | х | Х | х | х | х | х | Х | х | Reverse Cumulative Distribution Curves at Day 208 for ELISA Study Group 1 and 2: Percentage of Subjects vs. OspA ST3 Specific IgG Titer (GMT) by Age Cohort ([Booster] Per-Protocol Analysis Set) | |
| 60 | х | х | Х | х | х | х | x | х | х | Reverse Cumulative Distribution Curves at Day 208 for ELISA Study Group 1 and 2: Percentage of Subjects vs. OspA ST4 Specific IgG Titer (GMT) by Age Cohort ([Booster] Per-Protocol Analysis Set) | |
| 61 | x | х | х | х | х | х | х | Х | х | Reverse Cumulative Distribution Curves at Day 208 for ELISA Study Group 1 and 2: Percentage of Subjects vs. OspA ST5 Specific IgG Titer (GMT) by Age Cohort ([Booster] Per-Protocol Analysis Set) | |
| 62 | х | х | Х | х | х | х | х | х | х | Reverse Cumulative Distribution Curves at Day 208 for ELISA Study Group 1 and 2: Percentage of Subjects vs. OspA ST6 Specific IgG Titer (GMT) by Age Cohort ([Booster] Per-Protocol Analysis Set) | |
| 63 | | | Х | Х | х | х | х | Х | х | Reverse Cumulative Distribution Curves at Day 365 for ELISA Study Group 1 and 2: Percentage of Subjects vs. OspA ST1 Specific IgG Titer (GMT) by Age Cohort ([Booster] Per-Protocol Analysis Set) | |
| 64 | | | Х | Х | х | х | Х | Х | х | Reverse Cumulative Distribution Curves at Day 365 for ELISA Study Group 1 and 2: Percentage of Subjects vs. OspA ST2 Specific IgG Titer (GMT) by Age Cohort ([Booster] Per-Protocol Analysis Set) | |
| 65 | | | Х | х | х | х | х | х | х | Reverse Cumulative Distribution Curves at Day 365 for ELISA Study Group 1 and 2: Percentage of Subjects vs. OspA ST3 Specific IgG Titer (GMT) by Age Cohort ([Booster] Per-Protocol Analysis Set) | |
| 66 | | | х | х | х | х | х | х | х | Reverse Cumulative Distribution Curves at Day 365 for ELISA Study Group 1 and 2: Percentage of Subjects vs. OspA ST4 Specific IgG Titer (GMT) by Age Cohort ([Booster] Per-Protocol Analysis Set) | |
| 67 | | | Х | х | Х | х | Х | Х | х | Reverse Cumulative Distribution Curves at Day 365 for ELISA Study Group 1 and 2: Percentage of Subjects vs. OspA ST5 Specific IgG Titer (GMT) by Age Cohort ([Booster] Per-Protocol Analysis Set) | |

| | | | | Ar | nalysis | | | | | Figure Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Part | Α. | | | | Part E | 3 | | | Overall and |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4<br>3 | A5 | A6 | A7 | Legend | by age<br>cohort <sup>5</sup> |
| 68 | | | Х | х | х | х | Х | х | х | Reverse Cumulative Distribution Curves at Day 365 for ELISA Study Group 1 and 2: Percentage of Subjects vs. OspA ST6 Specific IgG Titer (GMT) by Age Cohort ([Booster] Per-Protocol Analysis Set) | |
| 69 | х | Х | Х | Х | х | Х | х | х | Х | Scatterplot: ELISA OspA ST1 Specific IgG Titer vs. ELISA OspA ST2 Specific IgG Titer at Day 208 for Pooled VLA15 Groups ([Booster] Per-Protocol Analysis Set) | |
| 70 | х | Х | Х | Х | х | Х | х | х | Х | Scatterplot: ELISA OspA ST1 Specific IgG Titer vs. ELISA OspA ST3 Specific IgG Titer at Day 208 for Pooled VLA15 Groups ([Booster] Per-Protocol Analysis Set) | |
| 71 | х | Х | х | Х | х | х | х | х | Х | Scatterplot: ELISA OspA ST1 Specific IgG Titer vs. ELISA OspA ST4 Specific IgG Titer at Day 208 for Pooled VLA15 Groups ([Booster] Per-Protocol Analysis Set) | |
| 72 | х | Х | х | х | х | х | х | х | Х | Scatterplot: ELISA OspA ST1 Specific IgG Titer vs. ELISA OspA ST5 Specific IgG Titer at Day 208 for Pooled VLA15 Groups ([Booster] Per-Protocol Analysis Set) | |
| 73 | Х | Х | Х | Х | х | Х | х | х | Х | Scatterplot: ELISA OspA ST1 Specific IgG Titer vs. ELISA OspA ST6 Specific IgG Titer at Day 208 for Pooled VLA15 Groups ([Booster] Per-Protocol Analysis Set) | |
| 74 | Х | Х | Х | Х | х | Х | х | х | Х | Scatterplot: ELISA OspA ST2 Specific IgG Titer vs. ELISA OspA ST3 Specific IgG Titer at Day 208 for Pooled VLA15 Groups ([Booster] Per-Protocol Analysis Set) | |
| 75 | х | Х | Х | Х | х | Х | х | х | Х | Scatterplot: ELISA OspA ST2 Specific IgG Titer vs. ELISA OspA ST4 Specific IgG Titer at Day 208 for Pooled VLA15 Groups ([Booster] Per-Protocol Analysis Set) | |
| 76 | х | х | х | Х | х | х | х | х | Х | Scatterplot: ELISA OspA ST2 Specific IgG Titer vs. ELISA OspA ST5 Specific IgG Titer at Day 208 for Pooled VLA15 Groups ([Booster] Per-Protocol Analysis Set) | |
| 77 | х | х | х | Х | х | х | х | х | Х | Scatterplot: ELISA OspA ST2 Specific IgG Titer vs. ELISA OspA ST6 Specific IgG Titer at Day 208 for Pooled VLA15 Groups ([Booster] Per-Protocol Analysis Set) | |
| 78 | х | х | х | Х | х | х | х | х | Х | Scatterplot: ELISA OspA ST3 Specific IgG Titer vs. ELISA OspA ST4 Specific IgG Titer at Day 208 for Pooled VLA15 Groups ([Booster] Per-Protocol Analysis Set) | |
| 79 | х | х | х | Х | х | х | х | х | Х | Scatterplot: ELISA OspA ST3 Specific IgG Titer vs. ELISA OspA ST5 Specific IgG Titer at Day 208 for Pooled VLA15 Groups ([Booster] Per-Protocol Analysis Set) | |
| 80 | х | Х | Х | Х | х | Х | х | х | Х | Scatterplot: ELISA OspA ST3 Specific IgG Titer vs. ELISA OspA ST6 Specific IgG Titer at Day 208 for Pooled VLA15 Groups ([Booster] Per-Protocol Analysis Set) | |
| 81 | х | х | Х | х | х | Х | х | х | Х | Scatterplot: ELISA OspA ST4 Specific IgG Titer vs. ELISA OspA ST5 Specific IgG Titer at Day 208 for Pooled VLA15 Groups ([Booster] Per-Protocol Analysis Set) | |
| 82 | Х | х | х | х | х | х | х | Х | х | Scatterplot: ELISA OspA ST4 Specific IgG Titer vs. ELISA OspA ST6 Specific IgG Titer at Day 208 for Pooled VLA15 Groups ([Booster] Per-Protocol Analysis Set) | |

| | Analysis | | | | | | | | | Figure Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Part | Α | | | | Part B | 3 | | | Overall and |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4<br>3 | A5 | A6 | A7 | Legend | by age<br>cohort <sup>5</sup> |
| 83 | х | Х | х | Х | Х | х | х | X | Х | Scatterplot: ELISA OspA ST5 Specific IgG Titer vs. ELISA OspA ST6 Specific IgG Titer at Day 208 for Pooled VLA15 Groups ([Booster] Per-Protocol Analysis Set) | |
| 84 | | | | | х | х | х | х | Х | Scatterplot: ELISA OspA ST1 Specific IgG Titer vs. ELISA OspA ST2 Specific IgG Titer at Month 19 for Pooled VLA15 Groups (Booster Per-Protocol Analysis Set) | |
| 85 | | | | | х | х | х | х | х | Scatterplot: ELISA OspA ST1 Specific IgG Titer vs. ELISA OspA ST3 Specific IgG Titer at Month 19 for Pooled VLA15 Groups (Booster Per-Protocol Analysis Set) | |
| 86 | | | | | х | х | х | х | Х | Scatterplot: ELISA OspA ST1 Specific IgG Titer vs. ELISA OspA ST4 Specific IgG Titer at Month 19 for Pooled VLA15 Groups (Booster Per-Protocol Analysis Set) | |
| 87 | | | | | Х | Х | х | Х | Х | Scatterplot: ELISA OspA ST1 Specific IgG Titer vs. ELISA OspA ST5 Specific IgG Titer at Month 19 for Pooled VLA15 Groups (Booster Per-Protocol Analysis Set) | |
| 88 | | | | | х | х | х | х | Х | Scatterplot: ELISA OspA ST1 Specific IgG Titer vs. ELISA OspA ST6 Specific IgG Titer at Month 19 for Pooled VLA15 Groups (Booster Per-Protocol Analysis Set) | |
| 89 | | | | | х | х | х | х | х | Scatterplot: ELISA OspA ST2 Specific IgG Titer vs. ELISA OspA ST3 Specific IgG Titer at Month 19 for Pooled VLA15 Groups (Booster Per-Protocol Analysis Set) | |
| 90 | | | | | х | х | х | х | х | Scatterplot: ELISA OspA ST2 Specific IgG Titer vs. ELISA OspA ST4 Specific IgG Titer at Month 19 for Pooled VLA15 Groups (Booster Per-Protocol Analysis Set) | |
| 91 | | | | | х | х | х | х | х | Scatterplot: ELISA OspA ST2 Specific IgG Titer vs. ELISA OspA ST5 Specific IgG Titer at Month 19 for Pooled VLA15 Groups (Booster Per-Protocol Analysis Set) | |
| 92 | | | | | х | х | х | Х | х | Scatterplot: ELISA OspA ST2 Specific IgG Titer vs. ELISA OspA ST6 Specific IgG Titer at Month 19 for Pooled VLA15 Groups (Booster Per-Protocol Analysis Set) | |
| 93 | | | | | х | х | х | х | х | Scatterplot: ELISA OspA ST3 Specific IgG Titer vs. ELISA OspA ST4 Specific IgG Titer at Month 19 for Pooled VLA15 Groups (Booster Per-Protocol Analysis Set) | |
| 94 | | | | | х | х | х | х | х | Scatterplot: ELISA OspA ST3 Specific IgG Titer vs. ELISA OspA ST5 Specific IgG Titer at Month 19 for Pooled VLA15 Groups (Booster Per-Protocol Analysis Set) | |
| 95 | | | | | х | х | х | х | х | Scatterplot: ELISA OspA ST3 Specific IgG Titer vs. ELISA OspA ST6 Specific IgG Titer at Month 19 for Pooled VLA15 Groups (Booster Per-Protocol Analysis Set) | |
| 96 | | | | | х | х | х | Х | Х | Scatterplot: ELISA OspA ST4 Specific IgG Titer vs. ELISA OspA ST5 Specific IgG Titer at Month 19 for Pooled VLA15 Groups (Booster] Per-Protocol Analysis Set) | |
| 97 | | | | | х | х | х | Х | Х | Scatterplot: ELISA OspA ST4 Specific IgG Titer vs. ELISA OspA ST6 Specific IgG Titer at Month 19 for Pooled VLA15 Groups (Booster Per-Protocol Analysis Set) | |
| 98 | | | | | х | Х | Х | Х | х | Scatterplot: ELISA OspA ST5 Specific IgG Titer vs. ELISA OspA ST6 Specific IgG Titer at Month 19 for Pooled VLA15 Groups (Booster Per-Protocol Analysis Set) | |




Adapted from:
STAT03\_A Statistical Analysis Plan

without prior written consent of




















#### 7.3.2 Adverse Events

| | | | | Aı | nalysis | | | | | Figure Description | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Part | t A | , | | | Part B | , | , | | Overall |
| ID | A1.1<br>A1.2<br>A1.3 | A1 | A2 | A3.1 | A3.2 | A4 | A5 | A6 | A7 | Legend | and by<br>age<br>cohort <sup>5</sup> |
| 1 | x | х | | | х | | | | | Bar Chart for Rate of Subjects with Solicited Local Adverse Events after any Vaccination by Symptom and Maximum Severity ([Booster] Safety Analysis Set) | х |
| 2 | х | х | | | х | | | | | Bar Chart for Rate of Subjects with Solicited Local Adverse Events Reaching FDA Toxicity Grading Scale after any Vaccination by Symptom and Maximum Severity ([Booster] Safety Analysis Set) | х |
| 3 | x | х | | | х | | | | | Bar Chart for Rate of Subjects with Solicited Local Adverse Events by Symptom, Maximum Severity and Vaccination Period ([Booster] Safety Analysis Set) | Х |
| 4 | х | х | | | х | | | | | Bar Chart for Rate of Subjects with Solicited Systemic Adverse Events after any Vaccination by Symptom and Maximum Severity ([Booster] Safety Analysis Set) | Х |
| 5 | х | Х | | | х | | | | | Bar Chart for Rate of Subjects with Solicited Systemic Adverse Events by Symptom, Maximum Severity and Vaccination Period ([Booster] Safety Analysis Set) | х |

### 8. SHELLS OF TABLES, DATA LISTINGS AND FIGURES

For this analysis, no table shells or mock tables will be produced, but analysis drafts of TLFs might be generated based on dummy group allocation (dummy randomization list) and dummy immunogenicity data. These drafts are reviewed by the sponsor prior to SAP finalization and database snapshot.

Adapted from: